CLINICAL TRIAL: NCT02332590
Title: A Randomized, Double-blind, Parallel-group Study Assessing the Efficacy and Safety of Sarilumab Monotherapy Versus Adalimumab Monotherapy in Patients With Rheumatoid Arthritis
Brief Title: Efficacy and Safety of Sarilumab and Adalimumab Monotherapy in Patients With Rheumatoid Arthritis (SARIL-RA-MONARCH)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC14092; 2014-002541-22 (EudraCT Number); U1111-1160-6154 (Other: UTN)
Record Dates: First submitted 2015-01-05; First posted 2015-01-07 (Estimated); Results first posted 2017-07-25 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — sarilumab; Adalimumab

STUDY DESIGN:
Intervention Model Description: During the OLE period of this study, all participants received sarilumab 200 mg or 150 mg q2w via prefilled syringe.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Adalimumab 40 mg/Sarilumab 200 mg (Active Comparator): Adalimumab 40 milligrams (mg) subcutaneous (SC) injection in combination with placebo for sarilumab every 2 weeks (q2w) for 24 weeks during the double-blind (DB) period. The dosing frequency of adalimumab was adjusted to 40 mg every week (qw) dosing in case of participants with inadequate response (less than [<] 20% improvement from baseline in tender joint count [TJC] and swollen joint count [SJC] for 2 consecutive visits) at or after Week 16 until Week 23. Participants who completed 24 weeks in the DB period had the option to continue in open label extension (OLE) period and received sarilumab 200 mg q2w until commercial availability of sarilumab in their country or up to a maximum of an additional 276 weeks (i.e. up to Week 300).
  Interventions: Drug: Adalimumab; Drug: Placebo (for sarilumab)
- Sarilumab 200 mg/Sarilumab 200 mg (Experimental): Sarilumab 200 mg SC injection in combination with placebo for adalimumab q2w for 24 weeks during the DB period. The dosing frequency of placebo for adalimumab was adjusted to 40 mg qw dosing in case of participants with inadequate response (<20% improvement from baseline in TJC and SJC for 2 consecutive visits) at or after Week 16 until Week 23. Participants who completed 24 weeks in the DB period had the option to continue in OLE period and received sarilumab 200 mg q2w until commercial availability of sarilumab in their country or up to a maximum of an additional 276 weeks (i.e. up to Week 300).
  Interventions: Drug: Sarilumab; Drug: Placebo (for adalimumab)

INTERVENTIONS:
Drug: Sarilumab — Pharmaceutical form: solution for injection in pre-filled syringe; Route of administration: SC
  Other Names: SAR153191; REGN88
  Arms: Sarilumab 200 mg/Sarilumab 200 mg
Drug: Adalimumab — Pharmaceutical form: solution for injection in pre-filled syringe; Route of administration: SC
  Other Names: Humira
  Arms: Adalimumab 40 mg/Sarilumab 200 mg
Drug: Placebo (for sarilumab) — Pharmaceutical form: solution for injection in pre-filled syringe; Route of administration: SC
  Arms: Adalimumab 40 mg/Sarilumab 200 mg
Drug: Placebo (for adalimumab) — Pharmaceutical form: solution for injection in pre-filled syringe; Route of administration: SC
  Arms: Sarilumab 200 mg/Sarilumab 200 mg

SUMMARY:
Primary Objective:

To demonstrate that sarilumab monotherapy was superior to adalimumab monotherapy with respect to signs and symptoms as assessed by disease activity score 28 (DAS28)-erythrocyte sedimentation rate (ESR) in participants with active rheumatoid arthritis (RA) who were either intolerant of, or considered inappropriate candidates for continued treatment with methotrexate (MTX), or after at least 12 weeks of continued treatment with MTX, were determined to be inadequate responders.

Secondary Objectives:

To demonstrate that sarilumab monotherapy was superior to adalimumab monotherapy in participants with active RA who were either intolerant of, or considered inappropriate candidates for continued treatment with MTX, or after at least 12 weeks of continued treatment with MTX, were determined to be inadequate responders, with respect to:

* Reduction of signs and symptoms of RA.
* Improvement in quality of life assessed by participant reported outcome questionnaires.

Assessment of the safety and tolerability of sarilumab monotherapy (including immunogenicity) throughout the study.

DETAILED DESCRIPTION:
Total study duration was up to 310 weeks: Up to a 4 week screening period, 24 week randomized double-blind treatment phase, 276-week open-label extension, and 6 weeks post-treatment final study visit.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of RA greater than or equal to (>=)3 months duration.
* American College of Rheumatology (ACR) Class I-III functional status.
* Active RA was defined as:

At least 6 of 66 swollen joints and 8 of 68 tender joints, high sensitivity C-reactive protein (hs-CRP) >=8 mg/L or ESR >=28 millimeter per hour (mm/H), and DAS28-ESR greater than (>) 5.1.

* Participants as per Investigator judgment were either intolerant of, or considered inappropriate candidates for continued treatment with MTX, or after at least 12 weeks of continued treatment with MTX, or inadequate responders treated with an adequate MTX dose for at least 12 weeks.

Exclusion criteria:

* Age <18 years or the legal age of consent in the country of the study site, whichever was higher.
* Current treatment with disease-modifying antirheumatic drug (DMARDs)/immunosuppressive agents including MTX, cyclosporine, mycophenolate, tacrolimus, gold, penicillamine, sulfasalazine or hydroxychloroquine within 2 weeks prior to the baseline (Randomization Visit) or azathioprine, cyclophosphamide within 12 weeks prior to baseline (Randomization Visit) or leflunomide within 8 weeks prior to the Randomization Visit, or 4 weeks after cholestyramine washout.
* Treatment with any prior biologic agent, including anti-interleukin 6 (IL-6), IL-6 receptor (IL-6R) antagonists, and prior treatment with a Janus kinase inhibitor.
* Use of parenteral corticosteroids or intra-articular corticosteroids within 4 weeks prior to screening.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 369 (Actual)
Dates: Start 2015-01-28 (Actual); Primary Completion 2016-01-20 (Actual); Study Completion 2020-12-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (86):
- United States (17):
  - Investigational Site Number 840407, Covina, California
  - Investigational Site Number 840400, Long Beach, California
  - Investigational Site Number 840141, Whittier, California
  - Investigational Site Number 840130, Lewes, Delaware
  - Investigational Site Number 840229, Coral Gables, Florida
  - Investigational Site Number 840128, Ormond Beach, Florida
  - Investigational Site Number 840403, St. Petersburg, Florida
  - Investigational Site Number 840140, Tampa, Florida
  - Investigational Site Number 840073, Cumberland, Maryland
  - Investigational Site Number 840202, Hagerstown, Maryland
  - Investigational Site Number 840232, Flint, Michigan
  - Investigational Site Number 840112, Lincoln, Nebraska
  - Investigational Site Number 840402, Charlotte, North Carolina
  - Investigational Site Number 840406, Hickory, North Carolina
  - Investigational Site Number 840404, Middleburg Heights, Ohio
  - Investigational Site Number 840127, Oklahoma City, Oklahoma
  - Investigational Site Number 840074, Mesquite, Texas
- Chile (7):
  - Investigational Site Number 152005, Osorno
  - Investigational Site Number 152001, Puerto Varas
  - Investigational Site Number 152002, Santiago
  - Investigational Site Number 152050, Santiago
  - Investigational Site Number 152014, Talca
  - Investigational Site Number 152015, Temuco IX Region
  - Investigational Site Number 152007, Viña del Mar
- Czechia (4):
  - Investigational Site Number 203001, Prague
  - Investigational Site Number 203033, Prague
  - Investigational Site Number 203030, Prague
  - Investigational Site Number 203002, Uherské Hradiště
- Germany (2):
  - Investigational Site Number 276058, Cologne
  - Investigational Site Number 276021, Osnabrück
- Hungary (5):
  - Investigational Site Number 348025, Budapest
  - Investigational Site Number 348020, Budapest
  - Investigational Site Number 348022, Budapest
  - Investigational Site Number 348024, Szombathely
  - Investigational Site Number 348023, Veszprém
- Israel (4):
  - Investigational Site Number 376032, Ashkelon
  - Investigational Site Number 376031, Haifa
  - Investigational Site Number 376030, Ramat Gan
  - Investigational Site Number 376011, Tel Aviv
- Peru (3):
  - Investigational Site Number 604003, Lima
  - Investigational Site Number 604005, Lima
  - Investigational Site Number 604022, Lima
- Poland (9):
  - Investigational Site Number 616056, Bytom
  - Investigational Site Number 616015, Elblag
  - Investigational Site Number 616005, Lublin
  - Investigational Site Number 616030, Lublin
  - Investigational Site Number 616055, Nadarzyn
  - Investigational Site Number 616018, Poznan
  - Investigational Site Number 616016, Szczecin
  - Investigational Site Number 616004, Warsaw
  - Investigational Site Number 616031, Warsaw
- Romania (5):
  - Investigational Site Number 642006, Brăila
  - Investigational Site Number 642001, Bucharest
  - Investigational Site Number 642010, Bucharest
  - Investigational Site Number 642002, Bucharest
  - Investigational Site Number 642005, Galati
- Russia (7):
  - Investigational Site Number 643006, Kemerovo
  - Investigational Site Number 643020, Moscow
  - Investigational Site Number 643001, Moscow
  - Investigational Site Number 643031, Moscow
  - Investigational Site Number 643030, Moscow
  - Investigational Site Number 643008, Saint Petersburg
  - Investigational Site Number 643011, Saratov
- South Africa (3):
  - Investigational Site Number 710011, Cape Town
  - Investigational Site Number 710007, Cape Town
  - Investigational Site Number 710004, Kempton Park
- South Korea (4):
  - Investigational Site Number 410005, Daegu
  - Investigational Site Number 410004, Daejeon
  - Investigational Site Number 410006, Seoul
  - Investigational Site Number 410001, Seoul
- Spain (6):
  - Investigational Site Number 724003, Barakaldo
  - Investigational Site Number 724015, Barcelona
  - Investigational Site Number 724011, Barcelona / Sabadell
  - Investigational Site Number 724001, Málaga
  - Investigational Site Number 724012, Santiago de Compostela
  - Investigational Site Number 724007, Seville
- Ukraine (9):
  - Investigational Site Number 804029, Ivano-Frankivsk
  - Investigational Site Number 804048, Kharkiv
  - Investigational Site Number 804014, Kyiv
  - Investigational Site Number 804047, Kyiv
  - Investigational Site Number 804037, Lutsk
  - Investigational Site Number 804046, Lviv
  - Investigational Site Number 804049, Poltava
  - Investigational Site Number 804011, Vinnitsya
  - Investigational Site Number 804043, Vinnitsya
- Investigational Site Number 826001, Leytonstone, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Burmester GR, Strand V, Kivitz AJ, Hu CC, Wang S, van Hoogstraten H, Klier GL, Fleischmann R. Long-term safety and efficacy of sarilumab with or without background csDMARDs in rheumatoid arthritis. Rheumatology (Oxford). 2023 Oct 3;62(10):3268-3279. doi: 10.1093/rheumatology/kead062. PMID 36727470
- [Derived] Choy E, Bykerk V, Lee YC, van Hoogstraten H, Ford K, Praestgaard A, Perrot S, Pope J, Sebba A. Disproportionate articular pain is a frequent phenomenon in rheumatoid arthritis and responds to treatment with sarilumab. Rheumatology (Oxford). 2023 Jul 5;62(7):2386-2393. doi: 10.1093/rheumatology/keac659. PMID 36413080
- [Derived] Rubbert-Roth A, Furst DE, Fiore S, Praestgaard A, Bykerk V, Bingham CO, Charles-Schoeman C, Burmester G. Association between low hemoglobin, clinical measures, and patient-reported outcomes in patients with rheumatoid arthritis: results from post hoc analyses of three phase III trials of sarilumab. Arthritis Res Ther. 2022 Aug 25;24(1):207. doi: 10.1186/s13075-022-02891-x. PMID 36008838
- [Derived] Rehberg M, Giegerich C, Praestgaard A, van Hoogstraten H, Iglesias-Rodriguez M, Curtis JR, Gottenberg JE, Schwarting A, Castaneda S, Rubbert-Roth A, Choy EHS; MOBILITY, MONARCH, TARGET, and ASCERTAIN investigators. Identification of a Rule to Predict Response to Sarilumab in Patients with Rheumatoid Arthritis Using Machine Learning and Clinical Trial Data. Rheumatol Ther. 2021 Dec;8(4):1661-1675. doi: 10.1007/s40744-021-00361-5. Epub 2021 Sep 14. PMID 34519964
- [Derived] Strand V, Boklage SH, Kimura T, Joly F, Boyapati A, Msihid J. High levels of interleukin-6 in patients with rheumatoid arthritis are associated with greater improvements in health-related quality of life for sarilumab compared with adalimumab. Arthritis Res Ther. 2020 Oct 20;22(1):250. doi: 10.1186/s13075-020-02344-3. PMID 33081825
- [Derived] Genovese MC, Burmester GR, Hagino O, Thangavelu K, Iglesias-Rodriguez M, John GS, Gonzalez-Gay MA, Mandrup-Poulsen T, Fleischmann R. Interleukin-6 receptor blockade or TNFalpha inhibition for reducing glycaemia in patients with RA and diabetes: post hoc analyses of three randomised, controlled trials. Arthritis Res Ther. 2020 Sep 9;22(1):206. doi: 10.1186/s13075-020-02229-5. PMID 32907617
- [Derived] Genovese MC, Fleischmann R, Kivitz A, Lee EB, van Hoogstraten H, Kimura T, St John G, Mangan EK, Burmester GR. Efficacy and safety of sarilumab in combination with csDMARDs or as monotherapy in subpopulations of patients with moderately to severely active rheumatoid arthritis in three phase III randomized, controlled studies. Arthritis Res Ther. 2020 Jun 10;22(1):139. doi: 10.1186/s13075-020-02194-z. PMID 32522251
- [Derived] Boyapati A, Schwartzman S, Msihid J, Choy E, Genovese MC, Burmester GR, Lam G, Kimura T, Sadeh J, Weinreich DM, Yancopoulos GD, Graham NMH. Association of High Serum Interleukin-6 Levels With Severe Progression of Rheumatoid Arthritis and Increased Treatment Response Differentiating Sarilumab From Adalimumab or Methotrexate in a Post Hoc Analysis. Arthritis Rheumatol. 2020 Sep;72(9):1456-1466. doi: 10.1002/art.41299. Epub 2020 Aug 25. PMID 32343882
- [Derived] Gabay C, Burmester GR, Strand V, Msihid J, Zilberstein M, Kimura T, van Hoogstraten H, Boklage SH, Sadeh J, Graham NMH, Boyapati A. Sarilumab and adalimumab differential effects on bone remodelling and cardiovascular risk biomarkers, and predictions of treatment outcomes. Arthritis Res Ther. 2020 Apr 7;22(1):70. doi: 10.1186/s13075-020-02163-6. PMID 32264972
- [Derived] Burmester GR, Strand V, Rubbert-Roth A, Amital H, Raskina T, Gomez-Centeno A, Pena-Rossi C, Gervitz L, Thangavelu K, St John G, Boklage S, Genovese MC. Safety and efficacy of switching from adalimumab to sarilumab in patients with rheumatoid arthritis in the ongoing MONARCH open-label extension. RMD Open. 2019 Oct 18;5(2):e001017. doi: 10.1136/rmdopen-2019-001017. eCollection 2019. PMID 31673415
- [Derived] Gossec L, Strand V, Proudfoot C, Chen CI, Guillonneau S, Kimura T, van Hoogstraten H, Mangan E, Reaney M. Effects of Sarilumab on Rheumatoid Arthritis as Reported by Patients Using the Rheumatoid Arthritis Impact of Disease Scale. J Rheumatol. 2019 Oct;46(10):1259-1267. doi: 10.3899/jrheum.180904. Epub 2019 Mar 15. PMID 30877216
- [Derived] Burmester GR, Lin Y, Patel R, van Adelsberg J, Mangan EK, Graham NM, van Hoogstraten H, Bauer D, Ignacio Vargas J, Lee EB. Efficacy and safety of sarilumab monotherapy versus adalimumab monotherapy for the treatment of patients with active rheumatoid arthritis (MONARCH): a randomised, double-blind, parallel-group phase III trial. Ann Rheum Dis. 2017 May;76(5):840-847. doi: 10.1136/annrheumdis-2016-210310. Epub 2016 Nov 17. PMID 27856432

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 86 centers in 15 countries. A total of 540 participants were involved in the study from 28 January 2015 to 29-December-2020, of whom 369 participants were randomized and 171 were screen failures. Screen failures were mainly due to exclusion criteria met and inclusion criteria not met.
Pre-assignment Details: Participants were randomized in 1:1 ratio (Adalimumab 40 milligrams (mg) every 2 weeks [q2w]: Sarilumab 200 mg q2w) and treated for 24 weeks in double-blind (DB) period of the study. Out of 321 participants who completed DB period, 320 participants entered the open label extension (OLE) period of the study.
Groups:
- Adalimumab 40 mg/Sarilumab 200 mg: Adalimumab 40 mg subcutaneous (SC) injection in combination with placebo for sarilumab q2w for 24 weeks during the DB period. The dosing frequency of adalimumab was adjusted to 40 mg every week (qw) dosing in case of participants with inadequate response (less than [<] 20% improvement from baseline in tender joint count [TJC] and swollen joint count [SJC] for 2 consecutive visits) at or after Week 16 until Week 23. Participants who completed 24 weeks in the DB period had the option to continue OLE period and received sarilumab 200 mg q2w until commercial availability of sarilumab in their country or up to a maximum of an additional 276 weeks (i.e. up to Week 300).
Period: DB Period (up to 24 Weeks)
Arm/Group | Adalimumab 40 mg/Sarilumab 200 mg | Sarilumab 200 mg/Sarilumab 200 mg
Started | 185 | 184
Treated | 184 | 184
Completed | 156 (155 participants entered OLE period and 1 did not enroll.) | 165
Not Completed | 29 | 19
Not completed — Adverse Event | 15 | 11
Not completed — Lack of Efficacy | 4 | 2
Not completed — Poor compliance to protocol | 3 | 1
Not completed — Randomized but not treated | 1 | 0
Not completed — Other than specified above | 6 | 5
Period: OLE Period (Week 24 up to Week 300)
Arm/Group | Adalimumab 40 mg/Sarilumab 200 mg | Sarilumab 200 mg/Sarilumab 200 mg
Started | 155 | 165
Completed | 108 | 120
Not Completed | 47 | 45
Not completed — Adverse Event | 20 | 23
Not completed — Lack of Efficacy | 2 | 6
Not completed — Poor compliance to protocol | 5 | 1
Not completed — Other Unspecified | 20 | 15

BASELINE CHARACTERISTICS:
Population: Analysis was performed on randomized population that included all participants who received at least 1 dose or part of a dose of Investigational Medicinal Product (IMP).
Groups:
- Adalimumab 40 mg/Sarilumab 200 mg: Adalimumab 40 mg SC injection in combination with placebo for sarilumab q2w for 24 weeks during the DB period. The dosing frequency of adalimumab was adjusted to 40 mg every week (qw) dosing in case of participants with inadequate response (< 20% improvement from baseline in TJC and SJC for 2 consecutive visits) at or after Week 16 until Week 23. Participants who completed 24 weeks in the DB period had the option to continue OLE period and received sarilumab 200 mg q2w until commercial availability of sarilumab in their country or up to a maximum of an additional 276 weeks (i.e. up to Week 300).
- Total: Total of all reporting groups
Arm/Group | Adalimumab 40 mg/Sarilumab 200 mg | Sarilumab 200 mg/Sarilumab 200 mg | Total
Number analyzed (Participants) | 185 | 184 | 369
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.6 (11.9) | 50.9 (12.6) | 52.2 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 150 | 157 | 307
  Male | 35 | 27 | 62
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian/White | 164 | 171 | 335
  Black | 3 | 1 | 4
  Asian/Oriental | 9 | 2 | 11
  Other | 9 | 10 | 19
Disease Activity Score 28 based on erythrocyte sedimentation rate (DAS28-ESR) [Mean (Standard Deviation); unit: units on a scale] — DAS28-ESR is a composite score that includes 4 variables: TJC (based on 28 joints); SJC (based on 28 joints); General health (GH) assessment by the participant assessed from the American College of Rheumatology (ACR) rheumatoid arthritis (RA) core set questionnaire (participant global assessment) in 100 mm visual analog scale (VAS); Marker of inflammation assessed by ESR in mm/hr.
  units on a scale | 6.76 (0.83) | 6.83 (0.76) | 6.80 (0.80)

OUTCOME MEASURES:

1. Primary Outcome: DB Period: Change From Baseline in Disease Activity Score for 28 Joints - Erythrocyte Sedimentation Rate (DAS28-ESR) Score at Week 24
Description: DAS28-ESR is a composite score that includes 4 variables: TJC (based on 28 joints); SJC (based on 28 joints); GH assessment by the participant assessed from the ACR and RA core set questionnaire (participant global assessment) in 100 mm VAS; Marker of inflammation assessed by ESR in mm/hr. The DAS28-ESR score provides a number indicating the current disease activity of the RA. DAS28-ESR total score ranges from 2-10. A DAS28-ESR score above 5.1 means high disease activity, DAS28-ESR score below 3.2 indicates low disease activity and DAS28-ESR score below 2.6 means disease remission. Least square (LS) mean and standard error (SE) at Week 24 were obtained using Mixed-effect model with repeated measures (MMRM) approach.
Time Frame: Baseline, Week 24
Population: Intent-to-treat (ITT) population included all participants. Overall Number of Participants Analyzed = participants with DAS28-ESR assessment at both baseline and Week 24.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Adalimumab 40 mg/Sarilumab 200 mg | Sarilumab 200 mg/Sarilumab 200 mg
Number analyzed (Participants) | 163 | 165
units on a scale | -2.20 (0.106) | -3.28 (0.105)
Statistical Analysis 1: Comparison: Adalimumab 40 mg/Sarilumab 200 mg vs Sarilumab 200 mg/Sarilumab 200 mg; Analysis was performed using MMRM approach with treatment, region, visits, and treatment-by-visit interaction as fixed effects and baseline DAS28-ESR score as a continuous covariate. Hierarchical testing procedure was used to control overall alpha error rate at 0.05 level and handle multiple endpoint analyses. Testing was then performed sequentially in order endpoints are reported. Hierarchical testing sequence continued only when previous endpoint was statistically significant at 0.05 level; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Threshold for significance at 0.05 level; LS Mean Difference = -1.077, 95% CI 2-sided [-1.361 to -0.793] — Sarilumab 200 mg vs. Adalimumab 40 mg

2. Secondary Outcome: DB Period: Percentage of Participants Achieving Clinical Remission Score (DAS28-ESR <2.6) at Week 24
Description: DAS28-ESR is a composite score that includes 4 variables: TJC (based on 28 joints); SJC (based on 28 joints); GH assessment by the participant assessed from the ACR RA core set questionnaire (participant global assessment) in 100 mm VAS; Marker of inflammation assessed by ESR in mm/hr. The DAS28-ESR score provides a number indicating the current disease activity of the RA. DAS28-ESR total score ranges from 2-10. A DAS28-ESR score above 5.1 means high disease activity, DAS28-ESR score below 3.2 indicates low disease activity and DAS28-ESR score below 2.6 means disease remission. Participants who discontinued treatment prior to Week 24 were analyzed as non-responders.
Time Frame: Week 24
Population: ITT Population.
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab 40 mg/Sarilumab 200 mg | Sarilumab 200 mg/Sarilumab 200 mg
Number analyzed (Participants) | 185 | 184
percentage of participants | 7.0 | 26.6
Statistical Analysis 1: Comparison: Adalimumab 40 mg/Sarilumab 200 mg vs Sarilumab 200 mg/Sarilumab 200 mg; Testing according to the hierarchical testing procedure (only performed if the previous endpoint was statistically significant). Analysis was performed using Cochran-Mantel-Haenszel method stratified by region; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance at 0.05 level; Odds Ratio (OR) = 4.879, 95% CI 2-sided [2.536 to 9.389] — Sarilumab 200 mg vs. Adalimumab 40 mg

3. Secondary Outcome: DB Period: Percentage of Participants Achieving ACR50 Criteria at Week 24
Description: ACR responses are assessed with a composite rating scale of the ACR that includes 7 variables: TJC (68 joints); SJC (66 joints); levels of an acute phase reactant (C-reactive protein [CRP] level); participant's assessment of pain (measured on 0 [no pain]-100 mm [worst pain] VAS); participant's global assessment of disease activity (measured on 0 [no arthritis activity]-100 mm [maximal arthritis activity] VAS); physician's global assessment of disease activity (measured on 0 [no arthritis activity]-100 mm [maximal arthritis activity] VAS); participant's assessment of physical function (measured by Health Assessment Questionnaire - Disability Index [HAQ-DI], with scoring range of 0 [better physical function] - 3 [worst physical function]). ACR50 is defined as achieving at least 50% improvement in both TJC and SJC, and at least 50% improvement in at least 3 of the 5 other assessments of the ACR. Participants were analyzed as non-responders from the time they discontinued treatment.
Time Frame: Week 24
Population: ITT Population.
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab 40 mg/Sarilumab 200 mg | Sarilumab 200 mg/Sarilumab 200 mg
Number analyzed (Participants) | 185 | 184
percentage of participants | 29.7 | 45.7
Statistical Analysis 1: Comparison: Adalimumab 40 mg/Sarilumab 200 mg vs Sarilumab 200 mg/Sarilumab 200 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0017, Cochran-Mantel-Haenszel — Threshold for significance at 0.05 level; Odds Ratio (OR) = 1.976, 95% CI 2-sided [1.289 to 3.028] — Sarilumab 200 mg vs. Adalimumab 40 mg

4. Secondary Outcome: DB Period: Percentage of Participants Achieving ACR70 Criteria at Week 24
Description: ACR responses are assessed with a composite rating scale of the ACR that includes 7 variables: TJC (68 joints); SJC (66 joints); levels of an acute phase reactant (CRP level); participant's assessment of pain (measured on 0 [no pain]-100 mm [worst pain] VAS); participant's global assessment of disease activity (measured on 0 [no arthritis activity]-100 mm [maximal arthritis activity] VAS); physician's global assessment of disease activity (measured on 0 [no arthritis activity]-100 mm [maximal arthritis activity] VAS); participant's assessment of physical function (measured by HAQ-DI, with scoring range of 0 [better physical function] - 3 [worst physical function]). ACR70 was defined as achieving at least 70% improvement in both TJC and SJC, and at least 70% improvement in at least 3 of the 5 other assessments. Participants were analyzed as non-responders from the time they discontinued treatment.
Time Frame: Week 24
Population: ITT Population.
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab 40 mg/Sarilumab 200 mg | Sarilumab 200 mg/Sarilumab 200 mg
Number analyzed (Participants) | 185 | 184
percentage of participants | 11.9 | 23.4
Statistical Analysis 1: Comparison: Adalimumab 40 mg/Sarilumab 200 mg vs Sarilumab 200 mg/Sarilumab 200 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0036, Cochran-Mantel-Haenszel — Threshold for significance at 0.05 level; Odds Ratio (OR) = 2.286, 95% CI 2-sided [1.300 to 4.020] — Sarilumab 200 mg vs. Adalimumab 40 mg

5. Secondary Outcome: DB Period: Percentage of Participants Achieving ACR20 Criteria at Week 24
Description: ACR responses are assessed with a composite rating scale of the ACR that includes 7 variables: TJC (68 joints); SJC (66 joints); levels of an acute phase reactant (CRP level); participant's assessment of pain (measured on 0 [no pain]-100 mm [worst pain] VAS); participant's global assessment of disease activity (measured on 0 [no arthritis activity]-100 mm [maximal arthritis activity] VAS); physician's global assessment of disease activity (measured on 0 [no arthritis activity]-100 mm [maximal arthritis activity] VAS); participant's assessment of physical function (measured by HAQ-DI, with scoring range of 0 [better physical function] - 3 [worst physical function]). ACR20 was defined as achieving at least 20% improvement in both TJC and SJC, and at least 20% improvement in at least 3 of the 5 other assessments. Participants were analyzed as non-responders from the time they discontinued treatment.
Time Frame: Week 24
Population: ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab 40 mg/Sarilumab 200 mg | Sarilumab 200 mg/Sarilumab 200 mg
Number analyzed (Participants) | 185 | 184
percentage of participants | 58.4 | 71.7
Statistical Analysis 1: Comparison: Adalimumab 40 mg/Sarilumab 200 mg vs Sarilumab 200 mg/Sarilumab 200 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0074, Cochran-Mantel-Haenszel — Threshold for significance 0.05 level; Odds Ratio (OR) = 1.800, 95% CI 2-sided [1.168 to 2.773] — Sarilumab 200 mg vs. Adalimumab 40 mg

6. Secondary Outcome: DB Period: Change From Baseline in HAQ-DI at Week 24
Description: Physical function was assessed by HAQ-DI. It consisted of at least 2 or 3 questions per category, participant reported assessment of ability to perform tasks in 8 categories of daily living activities: dress/groom; arise; eat; walk; reach; grip; hygiene; and common activities over past week rated on a 4-point scale where 0 = no difficulty; 1 = some difficulty; 2 = much difficulty; 3 = unable to do. Overall score was computed as the sum of category scores and divided by the number of categories answered, ranging from 0 to 3, where 0 = no disability and 3 = unable to do, high-dependency disability. LS mean and SE at Week 24 were obtained using MMRM approach.
Time Frame: Baseline, Week 24
Population: ITT population. Number of participants analyzed = participants with HAQ-DI assessment at both baseline and Week 24.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Adalimumab 40 mg/Sarilumab 200 mg | Sarilumab 200 mg/Sarilumab 200 mg
Number analyzed (Participants) | 158 | 165
units on a scale | -0.43 (0.045) | -0.61 (0.045)
Statistical Analysis 1: Comparison: Adalimumab 40 mg/Sarilumab 200 mg vs Sarilumab 200 mg/Sarilumab 200 mg; Testing according to the hierarchical testing procedure (only performed if the previous endpoint was statistically significant). Analysis was performed using MMRM approach with treatment, region, visits, and treatment-by-visit interaction as fixed effects and baseline HAQ-DI score as a continuous covariate; Test type: Superiority; p = 0.0037, Mixed Models Analysis — Threshold for significance at 0.05 level; LS Mean Difference = -0.182, 95% CI 2-sided [-0.305 to -0.059] — Sarilumab 200 mg vs. Adalimumab 40 mg

7. Secondary Outcome: DB Period: Change From Baseline in Short-Form-36 (SF-36) - Physical Component Summary (PCS) Score at Week 24
Description: SF-36 is a generic 36-item questionnaire consisting of 8 sub-scales, measures health-related quality of life (HRQL) in the last 4 weeks covering 2 summary measures: PCS and mental component summary (MCS). PCS with 4 sub-scales: physical function, role limitations due to physical problems, pain, and general health perception; and MCS with 4 sub-scales: vitality, social function, role limitations due to emotional problems, and mental health. Participants self-report on items in a sub-scale that have between 2-6 choices per item using Likert-type responses (e.g. none of the time, some of the time, etc.). Summations of item scores of the same sub-scale give the sub-scale scores, which are transformed into a range from 0 to 100; 0= worst HRQL, 100=best HRQL. Both PCS and MCS range from 0-100 with higher scores indicating better physical and mental health. LS mean and SE at Week 24 by MMRM approach.
Time Frame: Baseline, Week 24
Population: ITT population. Number of participants analyzed = participants with SF-36 PCS score assessment at both baseline and Week 24.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Adalimumab 40 mg/Sarilumab 200 mg | Sarilumab 200 mg/Sarilumab 200 mg
Number analyzed (Participants) | 157 | 159
units on a scale | 6.09 (0.555) | 8.74 (0.555)
Statistical Analysis 1: Comparison: Adalimumab 40 mg/Sarilumab 200 mg vs Sarilumab 200 mg/Sarilumab 200 mg; Testing according to the hierarchical testing procedure (only performed if the previous endpoint was statistically significant). Analysis was performed using MMRM approach with treatment, region, visits, and treatment-by-visit interaction as fixed effects and baseline SF-36 PCS score as a continuous covariate; Test type: Superiority; p = 0.0006, Mixed Models Analysis — Threshold for significance at 0.05 level; LS Mean Difference = 2.650, 95% CI 2-sided [1.147 to 4.153] — Sarilumab 200 mg vs. Adalimumab 40 mg

8. Secondary Outcome: DB Period: Change From Baseline in Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) Score at Week 24
Description: The FACIT-F is a 13-item questionnaire assessing fatigue where participants scored each item on a 5-point scale (0-4): 0=not at all, 1=a little bit, 2=somewhat, 3=quite a bit, 4=very much. A total score ranged from 0 to 52, where higher score corresponds to a lower level of fatigue. A positive change from baseline score indicates an improvement. LS mean and SE at Week 24 by MMRM approach.
Time Frame: Baseline, Week 24
Population: ITT population. Number of participants analyzed = participants with FACIT-F score assessment both at baseline and Week 24.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Adalimumab 40 mg/Sarilumab 200 mg | Sarilumab 200 mg/Sarilumab 200 mg
Number analyzed (Participants) | 158 | 165
units on a scale | 8.41 (0.709) | 10.18 (0.701)
Statistical Analysis 1: Comparison: Adalimumab 40 mg/Sarilumab 200 mg vs Sarilumab 200 mg/Sarilumab 200 mg; Testing according to the hierarchical testing procedure (only performed if the previous endpoint was statistically significant). Analysis was performed using MMRM approach with treatment, region, visits, and treatment-by-visit interaction as fixed effects and baseline FACIT-F score as a continuous covariate; Test type: Superiority; p = 0.0689, Mixed Models Analysis — Threshold for significance at 0.05 level; LS Mean Difference = 1.768, 95% CI 2-sided [-0.137 to 3.674] — Sarilumab 200 mg vs. Adalimumab 40 mg

9. Secondary Outcome: DB Period: Change From Baseline in SF-36 - Mental Health Component Summary Score at Week 24
Description: SF-36 is a generic 36-item questionnaire consisting of 8 sub-scales, measures HRQL in the last 4 weeks covering 2 summary measures: PCS and MCS. PCS with 4 subscales: physical function, role limitations due to physical problems, pain, and general health perception; and MCS with 4 subscales: vitality, social function, role limitations due to emotional problems, and mental health. Participants self-report on items in a subscale that have between 2-6 choices per item using Likert-type responses (e.g. none of the time, some of the time, etc.). Summations of item scores of the same sub-scale give the sub-scale scores, which are transformed into a range from 0 to 100; 0= worst HRQL, 100=best HRQL. Both PCS and MCS range from 0-100 with higher scores indicating better physical and mental health. LS mean and SE at Week 24 by MMRM approach.
Time Frame: Baseline, Week 24
Population: ITT population. Number of participants analyzed = participants with SF-36 - mental health component summary score assessment both at baseline and Week 24.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Adalimumab 40 mg/Sarilumab 200 mg | Sarilumab 200 mg/Sarilumab 200 mg
Number analyzed (Participants) | 157 | 159
units on a scale | 6.83 (0.774) | 7.86 (0.773)

10. Secondary Outcome: DB Period: Change From Baseline in Disease Activity Score for 28 Joints Based on C-Reactive Protein (DAS28-CRP Score) at Week 24
Description: DAS28-CRP is a composite score that includes 4 variables: TJC (based on 28 joints); SJC (based on 28 joints); GH assessment by the participant assessed from the ACR RA core set questionnaire (participant global assessment) in 100 mm VAS; Marker of inflammation assessed by high sensitivity C-reactive protein (hs-CRP) in mg/L. The DAS28-CRP score provides a number indicating the current disease activity of the RA. DAS28-CRP total score ranges from 2-10. A DAS28-CRP score above 5.1 means high disease activity, whereas a DAS28-CRP score below 3.2 indicates low disease activity and a DAS28-CRP score below 2.6 means disease remission. LS mean and SE at Week 24 were obtained using MMRM approach.
Time Frame: Baseline, Week 24
Population: ITT population. Number of participants analyzed = participants with DAS28-CRP score assessment at both baseline and Week 24.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Adalimumab 40 mg/Sarilumab 200 mg | Sarilumab 200 mg/Sarilumab 200 mg
Number analyzed (Participants) | 156 | 163
units on a scale | -1.97 (0.094) | -2.86 (0.093)

11. Secondary Outcome: DB Period: Percentage of Participants Achieving Clinical Remission Score (DAS28-CRP <2.6) at Week 24
Description: DAS28-CRP is a composite score that includes 4 variables: TJC (based on 28 joints); SJC (based on 28 joints); GH assessment by the participant assessed from the ACR RA core set questionnaire (participant global assessment) in 100 mm VAS; Marker of inflammation assessed by hs-CRP in mg/L. The DAS28-CRP score provides a number indicating the current disease activity of the RA. DAS28-CRP total score ranges from 2-10. A DAS28-CRP score above 5.1 means high disease activity, whereas a DAS28-CRP score below 3.2 indicates low disease activity and a DAS28-CRP score below 2.6 means disease remission. Participants were analyzed as non-responders from the time they discontinued treatment.
Time Frame: Week 24
Population: ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab 40 mg/Sarilumab 200 mg | Sarilumab 200 mg/Sarilumab 200 mg
Number analyzed (Participants) | 185 | 184
percentage of participants | 13.5 | 34.2

12. Secondary Outcome: DB Period: Percentage of Participants Achieving Low Disease Activity (DAS28-ESR < 3.2) at Week 24
Description: DAS28-ESR is a composite score that includes 4 variables: TJC (based on 28 joints); SJC (based on 28 joints); GH assessment by the participant assessed from the ACR RA core set questionnaire (participant global assessment) in 100 mm VAS; Marker of inflammation assessed by ESR in mm/hr. The DAS28-ESR score provides a number indicating the current disease activity of the RA. DAS28-ESR total score ranges from 2-10. A DAS28-ESR score above 5.1 means high disease activity, DAS28-ESR score below 3.2 indicates low disease activity and DAS28-ESR score below 2.6 means disease remission. Participants were analyzed as non-responders from the time they discontinued treatment.
Time Frame: Week 24
Population: ITT Population.
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab 40 mg/Sarilumab 200 mg | Sarilumab 200 mg/Sarilumab 200 mg
Number analyzed (Participants) | 185 | 184
percentage of participants | 14.1 | 42.9

13. Secondary Outcome: DB Period: Percentage of Participants Achieving Clinical Disease Activity Index (CDAI) Remission (CDAI ≤2.8) at Week 24
Description: CDAI is a composite index constructed to measure clinical remission in RA that does not include a laboratory test, and is a numerical summation of 4 components: SJC (28 joints), TJC (28 joints), participant's global assessment of disease activity (in cm), and physician's global assessment of disease activity (in cm). Total score ranges from 0 to 76 with a lower score indicating less disease activity. Participants were analyzed as non-responders from the time they discontinued treatment.
Time Frame: Week 24
Population: ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab 40 mg/Sarilumab 200 mg | Sarilumab 200 mg/Sarilumab 200 mg
Number analyzed (Participants) | 185 | 184
percentage of participants | 2.7 | 7.1

14. Secondary Outcome: DB Period: Change From Baseline in CDAI at Week 24
Description: CDAI is a composite index constructed to measure clinical remission in RA that does not include a laboratory test, and is a numerical summation of 4 components: SJC (28 joints), TJC (28 joints), participant's global assessment of disease activity (in cm), and physician's global assessment of disease activity (VAS in cm). Total score ranges from 0 to 76 with a lower score indicating less disease activity. A negative change in CDAI score indicates an improvement in disease activity and a positive change in score indicates a worsening of disease activity. LS means and SE at Week 24 were obtained using MMRM approach.
Time Frame: Baseline, Week 24
Population: ITT population. Number of participants analyzed = participants with CDAI assessment both at baseline and Week 24.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Adalimumab 40 mg/Sarilumab 200 mg | Sarilumab 200 mg/Sarilumab 200 mg
Number analyzed (Participants) | 158 | 165
units on a scale | -25.20 (0.842) | -28.94 (0.834)

15. Secondary Outcome: DB Period: Change From Baseline in European Quality of Life-5 Dimension 3 Level (EQ-5D-3L) Scores at Week 24
Description: EQ-5D-3L is a standardized, generic measure of health outcome. EQ-5D was designed for self-completion by participants. EQ-5D was specifically included to address concerns regarding the health economic impact of RA. EQ-5D-3L comprises of 5 questions on mobility, self-care, pain/discomfort, usual activities, and psychological status with 3 possible answers for each item (1=no problem, 2=moderate problems, 3=severe problems). The 5-dimensional 3-level systems are converted into a single index utility score between 0 to 1, where higher score indicates a better health state. EQ-5D-3L-VAS records the participant's self-rated health on a vertical VAS that allows the participants to indicate their health state that can range from 0 (worst imaginable) to 100 (best imaginable). LS mean and SE at Week 24 were obtained using MMRM approach.
Time Frame: Baseline, Week 24
Population: ITT population. Number of participants analyzed = participants with EQ-5D-3L score assessment both at baseline and Week 24. Here, Number Analyzed = participants with available data for specified category for each arm, respectively.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Adalimumab 40 mg/Sarilumab 200 mg | Sarilumab 200 mg/Sarilumab 200 mg
Number analyzed (Participants) | 156 | 164
units on a scale
  EQ-5D Single index utility score: number analyzed (Participants) | 156 | 160
  EQ-5D Single index utility score | 0.26 (0.019) | 0.32 (0.019)
  EQ-5D VAS | 19.94 (1.720) | 24.22 (1.686)

16. Secondary Outcome: DB Period: Change From Baseline in Rheumatoid Arthritis Impact of Disease (RAID) at Week 24
Description: RAID is a composite measure of the impact of RA on participants that takes into account 7 domains: pain, functional disability, fatigue, physical and emotional well-being, quality of sleep, and coping. The RAID is calculated based on 7 numerical rating scales (NRS) questions. Each NRS is assessed as a number between 0 and 10 that corresponds to the 7 domains. The values for each of these domains are weighed by participant assessment of relative importance and combined in a single score with a total score range of 0 (not affected, very good) to 10 (most affected). LS mean and SE at Week 24 were obtained using MMRM approach.
Time Frame: Baseline, Week 24
Population: ITT population. Number of participants analyzed = participants with RAID assessment both at baseline and Week 24.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Adalimumab 40 mg/Sarilumab 200 mg | Sarilumab 200 mg/Sarilumab 200 mg
Number analyzed (Participants) | 157 | 161
units on a scale | -2.30 (0.168) | -3.08 (0.168)

17. Secondary Outcome: DB Period: Change From Baseline in Work Productivity Survey - Rheumatoid Arthritis (WPS-RA) at Week 24: Work Days Missed Due to Arthritis
Description: The WPS-RA is a validated questionnaire that evaluates productivity limitations within work and within home associated with RA over the previous month. The questionnaire is interviewer-administered and based on participant self-report. It contains 9 questions addressing employment status (1 item), productivity at work (3 items), and within and outside the home (5 items). Number of work days missed in the last month by the participant was reported. LS mean and SE at Week 24 were obtained using MMRM approach.
Time Frame: Baseline, Week 24
Population: ITT population. Number of participants analyzed = participants with WPS-RA values available: Individual items assessment both at baseline and Week 24.
Measure: Least Squares Mean (Standard Error); unit: days
Arm/Group | Adalimumab 40 mg/Sarilumab 200 mg | Sarilumab 200 mg/Sarilumab 200 mg
Number analyzed (Participants) | 60 | 70
days | 0.05 (0.611) | -0.28 (0.547)

18. Secondary Outcome: DB Period: Change From Baseline in WPS-RA at Week 24: Days With Work Productivity Reduced by ≥ 50% Due to Arthritis
Description: The WPS-RA is a validated questionnaire that evaluates productivity limitations within work and within home associated with RA over the previous month. The questionnaire is interviewer-administered and based on participant self-report. It contains 9 questions addressing employment status (1 item), productivity at work (3 items), and within and outside the home (5 items). Number of work days with reduced productivity by >= 50% in the last month by the participants was reported. LS mean and SE at Week 24 were obtained using MMRM approach.
Time Frame: Baseline, Week 24
Population: as for outcome 17
Measure: Least Squares Mean (Standard Error); unit: days
Arm/Group | Adalimumab 40 mg/Sarilumab 200 mg | Sarilumab 200 mg/Sarilumab 200 mg
Number analyzed (Participants) | 60 | 70
days | -3.50 (0.525) | -3.74 (0.456)

19. Secondary Outcome: DB Period: Change From Baseline in WPS-RA at Week 24: Arthritis Interference With Work Productivity
Description: The WPS-RA is a validated questionnaire that evaluates productivity limitations within work and within home associated with RA over the previous month. The questionnaire is interviewer-administered and based on participant self-report. It contains 9 questions addressing employment status (1 item), productivity at work (3 items), and within and outside the home (5 items). Interference in the last month with work productivity was measured on a scale that ranges from 0 (no interference) to 10 (complete interference). LS mean and SE at Week 24 were obtained using MMRM approach.
Time Frame: Baseline, Week 24
Population: as for outcome 17
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Adalimumab 40 mg/Sarilumab 200 mg | Sarilumab 200 mg/Sarilumab 200 mg
Number analyzed (Participants) | 60 | 69
units on a scale | -2.510 (0.3470) | -2.919 (0.3073)

20. Secondary Outcome: DB Period: Change From Baseline in WPS-RA at Week 24: House Work Days Missed Due to Arthritis
Description: The WPS-RA is a validated questionnaire that evaluates productivity limitations within work and within home associated with RA over the previous month. The questionnaire is interviewer-administered and based on participant self-report. It contains 9 questions addressing employment status (1 item), productivity at work (3 items), and within and outside the home (5 items). Number of days with no household work in the last month by the participants was reported. LS mean and SE at Week 24 were obtained using MMRM approach.
Time Frame: Baseline, Week 24
Population: as for outcome 17
Measure: Least Squares Mean (Standard Error); unit: days
Arm/Group | Adalimumab 40 mg/Sarilumab 200 mg | Sarilumab 200 mg/Sarilumab 200 mg
Number analyzed (Participants) | 163 | 169
days | -4.22 (0.405) | -5.49 (0.400)

21. Secondary Outcome: DB Period: Change From Baseline in WPS-RA at Week 24: Days With Household Work Productivity Reduced by >= 50% Due to Arthritis
Description: The WPS-RA is a validated questionnaire that evaluates productivity limitations within work and within home associated with RA over the previous month. The questionnaire is interviewer-administered and based on participant self-report. It contains 9 questions addressing employment status (1 item), productivity at work (3 items), and within and outside the home (5 items). Number of days with reduced household work productivity by >= 50% in the last month by the participants was reported. LS mean and SE at Week 24 were obtained using MMRM approach.
Time Frame: Baseline, Week 24
Population: as for outcome 17
Measure: Least Squares Mean (Standard Error); unit: days
Arm/Group | Adalimumab 40 mg/Sarilumab 200 mg | Sarilumab 200 mg/Sarilumab 200 mg
Number analyzed (Participants) | 163 | 169
days | -4.87 (0.451) | -6.70 (0.445)

22. Secondary Outcome: DB Period: Change From Baseline in WPS-RA at Week 24: Days With Family/Social/Leisure Activities Missed Due to Arthritis
Description: The WPS-RA is a validated questionnaire that evaluates productivity limitations within work and within home associated with RA over the previous month. The questionnaire is interviewer-administered and based on participant self-report. It contains 9 questions addressing employment status (1 item), productivity at work (3 items), and within and outside the home (5 items). Number of days missed of family/social/leisure activities in the last month by the participants was reported. LS mean and SE at Week 24 were obtained using MMRM approach.
Time Frame: Baseline, Week 24
Population: as for outcome 17
Measure: Least Squares Mean (Standard Error); unit: days
Arm/Group | Adalimumab 40 mg/Sarilumab 200 mg | Sarilumab 200 mg/Sarilumab 200 mg
Number analyzed (Participants) | 163 | 169
days | -3.33 (0.376) | -4.14 (0.371)

23. Secondary Outcome: DB Period: Change From Baseline in WPS-RA at Week 24: Days With Outside Help Hired Due to Arthritis
Description: The WPS-RA is a validated questionnaire that evaluates productivity limitations within work and within home associated with RA over the previous month. The questionnaire is interviewer-administered and based on participant self-report. It contains 9 questions addressing employment status (1 item), productivity at work (3 items), and within and outside the home (5 items). Number of days with outside help hired in the last month by the participant was reported. LS mean and SE at Week 24 were obtained using MMRM approach.
Time Frame: Baseline, Week 24
Population: ITT population. Number of participants analyzed =participants with WPS-RA values available: Individual items assessment both at baseline and Week 24.
Measure: Least Squares Mean (Standard Error); unit: days
Arm/Group | Adalimumab 40 mg/Sarilumab 200 mg | Sarilumab 200 mg/Sarilumab 200 mg
Number analyzed (Participants) | 163 | 168
days | -2.57 (0.401) | -3.43 (0.398)

24. Secondary Outcome: DB Period: Change From Baseline in WPS-RA at Week 24: RA Interference With Household Work Productivity
Description: The WPS-RA is a validated questionnaire that evaluates productivity limitations within work and within home associated with RA over the previous month. The questionnaire is interviewer-administered and based on participant self-report. It contains 9 questions addressing employment status (1 item), productivity at work (3 items), and within and outside the home (5 items). The RA interference in the last month with household work productivity was measured on a scale that ranges from 0 (no interference) to 10 (complete interference). LS mean and SE at Week 24 were obtained using MMRM approach.
Time Frame: Baseline, Week 24
Population: as for outcome 17
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Adalimumab 40 mg/Sarilumab 200 mg | Sarilumab 200 mg/Sarilumab 200 mg
Number analyzed (Participants) | 163 | 168
units on a scale | -2.605 (0.2110) | -3.276 (0.2099)

25. Secondary Outcome: DB Period: Change From Baseline in Morning Stiffness VAS at Week 24
Description: RA is associated with stiffness of joints, especially in the morning after prolonged stationery state. The degree of stiffness can be an indicator of disease severity. The severity of morning stiffness was assessed on a VAS scale from 0 mm (no problem) to 100 mm (major problem). LS mean and SE at Week 24 were obtained using MMRM approach.
Time Frame: Baseline, Week 24
Population: ITT population. Number of participants analyzed = participants with morning stiffness VAS assessment both at baseline and Week 24.
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Adalimumab 40 mg/Sarilumab 200 mg | Sarilumab 200 mg/Sarilumab 200 mg
Number analyzed (Participants) | 156 | 165
mm | -29.29 (1.970) | -35.08 (1.947)

26. Secondary Outcome: DB Period: Change From Baseline in Individual ACR Component - TJC and SJC at Week 24
Description: ACR components were: TJC, SJC, physician global VAS, participant global VAS, pain VAS, HAQ-DI & acute phase reactant (hs-CRP and ESR levels). 68 joints were assessed for tenderness (TJC scoring 0-68) and 66 joints for swelling (SJC scoring 0-66). The 66 SJC evaluated the following joints: temporomandibular, sternoclavicular, acromioclavicular, shoulder, elbow, wrist, metacarpophalangeal, interphalangeal of thumb, distal interphalangeal, proximal interphalangeal, knee, ankle mortise, ankle tarsus, metatarsophalangeal, interphalangeal of great toe, and proximal/distal interphalangeal of the toes. The TJC examined hip joints, in addition to the joints assessed for SJC. Increase in number of tender joints/swollen joints indicated severity. LS mean and SE at Week 24 were obtained using MMRM approach.
Time Frame: Baseline, Week 24
Population: ITT population. Number of participants analyzed = participants with TJC and SJC assessment both at baseline and Week 24.
Measure: Least Squares Mean (Standard Error); unit: joints
Arm/Group | Adalimumab 40 mg/Sarilumab 200 mg | Sarilumab 200 mg/Sarilumab 200 mg
Number analyzed (Participants) | 158 | 166
joints
  TJC | -16.45 (0.781) | -18.23 (0.772)
  SJC | -12.20 (0.450) | -13.44 (0.444)

27. Secondary Outcome: DB Period: Change From Baseline in Individual ACR Component - Physician Global VAS, Participant Global VAS and Pain VAS at Week 24
Description: ACR components were: TJC, SJC, physician global VAS, participant global VAS, pain VAS, HAQ-DI & acute phase reactant (hs-CRP and ESR levels). Physician global VAS & participant global VAS was done on 100 mm horizontal anchored VAS, ranging from 0 "no arthritis activity" to 100 "maximal arthritis activity" and Pain VAS on 100 mm VAS, ranging from 0 "no pain" to 100 "worst pain". LS mean and SE at Week 24 were obtained using MMRM approach.
Time Frame: Baseline, Week 24
Population: ITT population. Number of participants analyzed = participants with individual ACR components assessment both at baseline and Week 24. Here, Number Analyzed = participants with available data for specified category for each arm, respectively.
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Adalimumab 40 mg/Sarilumab 200 mg | Sarilumab 200 mg/Sarilumab 200 mg
Number analyzed (Participants) | 158 | 166
mm
  Physician global VAS | -37.80 (1.431) | -45.33 (1.414)
  Participant global VAS: number analyzed (Participants) | 158 | 165
  Participant global VAS | -24.82 (1.752) | -33.30 (1.731)
  Pain VAS: number analyzed (Participants) | 157 | 165
  Pain VAS | -27.41 (1.802) | -36.19 (1.776)

28. Secondary Outcome: DB Period: Change From Baseline in Individual ACR Component - CRP Level at Week 24
Description: ACR components were: TJC, SJC, physician global VAS, participant global VAS, pain VAS, HAQ-DI & acute phase reactant (hs-CRP and ESR levels). An elevated CRP level is considered a non-specific "marker" for RA. A decrease indicates improvement. LS mean and SE at Week 24 were obtained using MMRM approach.
Time Frame: Baseline, Week 24
Population: ITT population. Number of participants analyzed = participants with CRP assessment both at baseline and Week 24.
Measure: Least Squares Mean (Standard Error); unit: mg/L
Arm/Group | Adalimumab 40 mg/Sarilumab 200 mg | Sarilumab 200 mg/Sarilumab 200 mg
Number analyzed (Participants) | 156 | 164
mg/L | -2.91 (1.461) | -17.01 (1.431)

29. Secondary Outcome: DB Period: Change From Baseline in Individual ACR Component- ESR Level at Week 24
Description: ACR components were: TJC, SJC, physician global VAS, participant global VAS, pain VAS, HAQ-DI & acute phase reactant (hs-CRP and ESR levels). The ESR is a blood test that can reveal inflammatory activity. Inflammation can cause the cells to clump together. The farther the red blood cells have descended, the greater the inflammatory response. LS mean and SE at Week 24 were obtained using MMRM approach.
Time Frame: Baseline, Week 24
Population: ITT population. Number of participants analyzed = participants with ESR assessment both at baseline and Week 24.
Measure: Least Squares Mean (Standard Error); unit: mm/hr
Arm/Group | Adalimumab 40 mg/Sarilumab 200 mg | Sarilumab 200 mg/Sarilumab 200 mg
Number analyzed (Participants) | 163 | 166
mm/hr | -12.74 (1.398) | -32.11 (1.388)

30. Secondary Outcome: DB Period: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: Adverse event (AE) was defined as any untoward medical occurrence in participant who received investigational medicinal product (IMP) and did not necessarily had to have causal relationship with treatment. All reported AEs are TEAEs developed/worsened during 'on treatment period' (time from first dose of study drug up to day before first dose of open-label treatment for participants who completed 24-week randomized//DB treatment). SAEs were AEs resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly or a medically important event.
Time Frame: From Week 0 to Week 24
Population: Analysis was performed on safety population (DB period) which consisted of all randomized participants who received at least one dose of study medication analyzed according to the treatment they have actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Adalimumab 40 mg/Sarilumab 200 mg | Sarilumab 200 mg/Sarilumab 200 mg
Number analyzed (Participants) | 184 | 184
Participants
  TEAEs | 117 | 118
  SAEs | 13 | 9

31. Secondary Outcome: OLE Period: Number of Participants With Treatment-emergent Adverse Events and Serious Adverse Events
Description: AE was defined as any untoward medical occurrence in participant who received IMP and did not necessarily had to have causal relationship with treatment. All reported AEs are TEAEs developed/worsened during 'on treatment period' (from end of week 24 [Baseline of OLE Period] up to last dose in OLE period + 6 weeks [follow-up], regardless of unplanned intermittent discontinuations). SAEs were AEs resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly or a medically important event.
Time Frame: From end of Week 24 (Baseline of OLE Period) up to last dose in OLE + 6 weeks of follow up (i.e. up to Week 306)
Population: Analysis was performed on safety population (OLE period) which included all randomized participants who continued OLE period and received at least one dose of the study medication during OLE period, analyzed according to the treatment they have actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Adalimumab 40 mg/Sarilumab 200 mg | Sarilumab 200 mg/Sarilumab 200 mg
Number analyzed (Participants) | 155 | 165
Participants
  TEAE | 135 | 143
  SAE | 31 | 25

32. Secondary Outcome: DB Period: Number of Participants With Potentially Clinically Significant Abnormalities (PCSA) - Hematological Parameters
Description: Criteria for potentially clinically significant laboratory abnormalities included:
  * Hemoglobin (Hb): less than or equal to (<=) 115 grams per liter (g/L) (Male), <= 95 g/L (Female); greater than or equal to (>=) 185 g/L (18.5 g/dL) (Male), >= 165 g/L (16.5 g/dL) (Female); Decrease From Baseline (DFB) = 20 g/L (2 g/dL).
  * Hematocrit: <= 0.37 volume/volume (v/v) (Male); <= 0.32 v/v (F); >= 0.55 v/v (Male); >= 0.5 v/v (Female).
  * Red Blood Cells (RBCs): >=6 Tera/ liter (L).
  * Platelets: < 50 Giga/L, 50 - 100 Giga/L, >= 700 Giga/L.
  * White blood cells (WBC): < 3.0 Giga/L (Non-Black); < 2.0 Giga/L (Black), >= 16.0 Giga/L.
  * Neutrophils: < 1.0 Giga/L, < 1.5 Giga/L (Non-Black); < 1.0 Giga/L (Black).
  * Lymphocytes: < 0.5 Giga/L, >= 0.5 Giga/L - lower limit of normal (LLN), > 4.0 Giga/L.
  * Monocytes: > 0.7 Giga/L.
  * Basophils: > 0.1 Giga/L.
  * Eosinophils: > 0.5 Giga/L or > upper limit of normal (ULN) (if ULN >= 0.5 Giga/L).
Time Frame: From Week 0 to Week 24
Population: Analysis was performed on safety population (DB Period). Here, 'number analyzed' = participants with available data for each specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | Adalimumab 40 mg/Sarilumab 200 mg | Sarilumab 200 mg/Sarilumab 200 mg
Number analyzed (Participants) | 184 | 184
Participants
  Hb:<=115 g/L, <=95 g/L | 12 | 7
  Hb: >=185 g/L, >=165 g/L | 0 | 1
  Hb: DFB >=20 g/L | 5 | 5
  Hematocrit: <= 0.37 v/v; <=0.32 v/v: number analyzed (Participants) | 183 | 184
  Hematocrit: <= 0.37 v/v; <=0.32 v/v | 21 | 10
  Hematocrit: >=0.55 v/v; >=0.5 v/v: number analyzed (Participants) | 183 | 184
  Hematocrit: >=0.55 v/v; >=0.5 v/v | 1 | 3
  RBCs: >=6 Tera/L | 0 | 1
  Platelets: < 50 Giga/L: number analyzed (Participants) | 183 | 184
  Platelets: < 50 Giga/L | 0 | 1
  Platelets: 50 - 100 Giga/L: number analyzed (Participants) | 183 | 184
  Platelets: 50 - 100 Giga/L | 0 | 0
  Platelets: >= 700 Giga/L: number analyzed (Participants) | 183 | 184
  Platelets: >= 700 Giga/L | 1 | 0
  WBC: < 3.0 Giga/L (Non-Black); < 2.0 Giga/L (Black) | 1 | 32
  WBC: >= 16.0 Giga/L | 8 | 5
  Neutrophils: < 1.0 Giga/L: number analyzed (Participants) | 183 | 184
  Neutrophils: < 1.0 Giga/L | 2 | 19
  Neutrophils: < 1.5 Giga/L (Non-Black); < 1.0 Giga/L (Black): number analyzed (Participants) | 183 | 184
  Neutrophils: < 1.5 Giga/L (Non-Black); < 1.0 Giga/L (Black) | 7 | 50
  Lymphocytes: < 0.5 Giga/L: number analyzed (Participants) | 183 | 184
  Lymphocytes: < 0.5 Giga/L | 2 | 2
  Lymphocytes: >= 0.5 Giga/L - LLN: number analyzed (Participants) | 183 | 184
  Lymphocytes: >= 0.5 Giga/L - LLN | 8 | 21
  Lymphocytes: > 4.0 Giga/L: number analyzed (Participants) | 183 | 184
  Lymphocytes: > 4.0 Giga/L | 17 | 6
  Monocytes: > 0.7 Giga/L: number analyzed (Participants) | 183 | 184
  Monocytes: > 0.7 Giga/L | 46 | 38
  Basophils: > 0.1 Giga/L: number analyzed (Participants) | 183 | 184
  Basophils: > 0.1 Giga/L | 53 | 37
  Eosinophils: > 0.5 Giga/L or > ULN (if ULN >= 0.5 Giga/L): number analyzed (Participants) | 183 | 184
  Eosinophils: > 0.5 Giga/L or > ULN (if ULN >= 0.5 Giga/L) | 4 | 9

33. Secondary Outcome: OLE Period: Number of Participants With Potentially Clinically Significant Abnormalities - Hematological Parameters
Description: Criteria for potentially clinically significant laboratory abnormalities included:
  * Hb: <=115 g/L (Male), <= 95 g/L (Female); >=185 g/L (18.5 g/dL) (Male), >= 165 g/L (16.5 g/dL) (Female); DFB >= 20 g/L (2 g/dL).
  * Hematocrit: <= 0.37 v/v (Male); <= 0.32 v/v (Female); >= 0.55 v/v (Male); >= 0.5 v/v (Female).
  * RBCs: >=6 Tera/ L.
  * Platelets: < 50 Giga/L, >=50 - 100 Giga/L, >= 700 Giga/L.
  * WBC: < 3.0 Giga/L (Non-Black); < 2.0 Giga/L (Black), >= 16.0 Giga/L.
  * Neutrophils: < 1.0 Giga/L, < 1.5 Giga/L (Non-Black); < 1.0 Giga/L (Black).
  * Lymphocytes: < 0.5 Giga/L, >= 0.5 Giga/L - LLN, > 4.0 Giga/L.
  * Monocytes: > 0.7 Giga/L.
  * Basophils: > 0.1 Giga/L.
  * Eosinophils: > 0.5 Giga/L or > ULN (if ULN >= 0.5 Giga/L).
Time Frame: From end of Week 24 (Baseline of OLE Period) up to Week 300
Population: Analysis was performed on safety population (OLE Period). Here, 'overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Adalimumab 40 mg/Sarilumab 200 mg | Sarilumab 200 mg/Sarilumab 200 mg
Number analyzed (Participants) | 154 | 165
Participants
  Hb:<=115 g/L, <=95 g/L | 8 | 5
  Hb: >=185 g/L, >=165 g/L | 3 | 3
  Hb: DFB >=20 g/L | 13 | 13
  Hematocrit: <= 0.37 v/v; <=0.32 v/v | 12 | 14
  Hematocrit: >=0.55 v/v; >=0.5 v/v | 5 | 8
  RBCs: >=6 Tera/L | 3 | 2
  Platelets: < 50 Giga/L | 0 | 0
  Platelets: >=50 - 100 Giga/L | 4 | 4
  Platelets: >= 700 Giga/L | 2 | 1
  WBC: < 3.0 Giga/L (Non-Black); < 2.0 Giga/L (Black) | 34 | 46
  WBC: >= 16.0 Giga/L | 11 | 7
  Neutrophils: < 1.0 Giga/L | 24 | 25
  Neutrophils: < 1.5 Giga/L (Non-Black); < 1.0 Giga/L (Black) | 62 | 69
  Lymphocytes: < 0.5 Giga/L | 2 | 3
  Lymphocytes: >= 0.5 Giga/L - LLN | 28 | 42
  Lymphocytes: > 4.0 Giga/L | 15 | 7
  Monocytes: > 0.7 Giga/L | 48 | 43
  Basophils: > 0.1 Giga/L | 78 | 70
  Eosinophils: > 0.5 Giga/L or > ULN (if ULN >= 0.5 Giga/L) | 11 | 14

34. Secondary Outcome: DB Period: Number of Participants With Potentially Clinically Significant Abnormalities - Liver Function Tests
Description: Criteria for potentially clinically significant abnormalities:
  * Alanine Aminotransferase (ALT): >1 ULN and <=1.5 ULN; >1.5 ULN and <=3 ULN; >3 ULN and <=5 ULN; >5 ULN and <=10 ULN; >10 ULN and <=20 ULN; >20 ULN.
  * Aspartate aminotransferase (AST): >1 ULN and <=1.5 ULN; >1.5 ULN and <=3 ULN; >3 ULN and <=5 ULN; >5 ULN and <=10 ULN; >10 ULN and <=20 ULN; >20 ULN.
  * Alkaline phosphatase: >1.5 ULN.
  * Total bilirubin (TBILI): >1.5 ULN; >2 ULN.
  * Conjugated bilirubin (CBILI): >1.5 ULN.
  * Unconjugated bilirubin: >1.5 ULN, >2 ULN.
  * ALT >3 ULN and TBILI >2 ULN.
  * CBILI >35% TBILI and TBILI >1.5 ULN.
  * Albumin: <=25 g/L.
Time Frame: From Week 0 to Week 24
Population: Analysis was performed on safety population (DB Period). Here, 'overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Adalimumab 40 mg/Sarilumab 200 mg | Sarilumab 200 mg/Sarilumab 200 mg
Number analyzed (Participants) | 183 | 184
Participants
  ALT >1 ULN and <=1.5 ULN | 22 | 36
  ALT >1.5 ULN and <=3 ULN | 17 | 26
  ALT >3 ULN and <=5 ULN | 3 | 5
  ALT >5 ULN and <=10 ULN | 1 | 1
  ALT >10 ULN and <=20 ULN | 1 | 0
  ALT >20 ULN | 0 | 0
  AST >1 ULN and <=1.5 ULN | 16 | 22
  AST >1.5 ULN and <=3 ULN | 7 | 13
  AST >3 ULN and <=5 ULN | 3 | 2
  AST >5 ULN and <=10 ULN | 0 | 0
  AST >10 ULN and <=20 ULN | 1 | 0
  AST >20 ULN | 0 | 0
  Alkaline Phosphatase >1.5 ULN | 6 | 2
  TBILI >1.5 ULN | 1 | 7
  TBILI >2 ULN | 0 | 2
  CBILI >1.5 ULN | 0 | 0
  Unconjugated Bilirubin >1.5 ULN | 5 | 13
  Unconjugated Bilirubin >2 ULN | 1 | 7
  ALT> 3 ULN and TBILI >2 ULN | 0 | 0
  CBILI >35% TBILI and TBILI >1.5 ULN | 0 | 0
  Albumin <=25 g/L | 0 | 0

35. Secondary Outcome: OLE Period: Number of Participants With Potentially Clinically Significant Abnormalities - Liver Function Tests
Description: Criteria for potentially clinically significant abnormalities:
  * ALT: >1 ULN and <=1.5 ULN; >1.5 ULN and <=3 ULN; >3 ULN and <=5 ULN; >5 ULN and <=10 ULN; >10 ULN and <=20 ULN; >20 ULN.
  * AST: >1 ULN and <=1.5 ULN; >1.5 ULN and <=3 ULN; >3 ULN and <=5 ULN; >5 ULN and <=10 ULN; >10 ULN and <=20 ULN; >20 ULN.
  * Alkaline phosphatase: >1.5 ULN.
  * TBILI: >1.5 ULN; >2 ULN.
  * CBILI: >1.5 ULN.
  * Unconjugated bilirubin: >1.5 ULN, >2 ULN.
  * ALT >3 ULN and TBILI >2 ULN.
  * CBILI >35% TBILI and TBILI >1.5 ULN.
  * Albumin: <=25 g/L.
Time Frame: From end of Week 24 (Baseline of OLE Period) up to Week 300
Population: as for outcome 33
Measure: Count of Participants; unit: Participants
Arm/Group | Adalimumab 40 mg/Sarilumab 200 mg | Sarilumab 200 mg/Sarilumab 200 mg
Number analyzed (Participants) | 154 | 165
Participants
  ALT >1 ULN and <=1.5 ULN | 41 | 36
  ALT >1.5 ULN and <=3 ULN | 31 | 34
  ALT >3 ULN and <=5 ULN | 11 | 10
  ALT >5 ULN and <=10 ULN | 1 | 6
  ALT >10 ULN and <=20 ULN | 0 | 2
  ALT >20 ULN | 1 | 1
  AST >1 ULN and <=1.5 ULN | 25 | 39
  AST >1.5 ULN and <=3 ULN | 23 | 17
  AST >3 ULN and <=5 ULN | 2 | 7
  AST >5 ULN and <=10 ULN | 2 | 2
  AST >10 ULN and <=20 ULN | 0 | 0
  AST >20 ULN | 0 | 1
  Alkaline Phosphatase >1.5 ULN | 0 | 1
  TBILI >1.5 ULN | 11 | 6
  TBILI >2 ULN | 3 | 1
  CBILI >1.5 ULN | 0 | 0
  Unconjugated Bilirubin >1.5 ULN | 21 | 22
  Unconjugated Bilirubin >2 ULN | 11 | 10
  ALT> 3 ULN and TBILI >2 ULN | 1 | 0
  CBILI >35% TBILI and TBILI >1.5 ULN | 0 | 0
  Albumin <=25 g/L | 0 | 0

36. Secondary Outcome: DB Period: Number of Participants With Potentially Clinically Significant Abnormalities - Metabolic Parameters
Description: Criteria for potentially clinically significant abnormalities:
  * Glucose: <=3.9 millimole/liter (mmol/L) and <LLN; >=11.1 mmol/L (unfasted [unfas]) or >=7 mmol/L (fasted [fas]).
  * Hemoglobin A1c (HbA1c): >8%.
  * Total cholesterol: >=6.2 mmol/L; >=7.74 mmol/L.
  * LDL cholesterol: >=4.1 mmol/L; >=4.9 mmol/L.
  * Triglycerides: >=4.6 mmol/L; >=5.6 mmol/L.
Time Frame: From Week 0 to Week 24
Population: as for outcome 32
Measure: Count of Participants; unit: Participants
Arm/Group | Adalimumab 40 mg/Sarilumab 200 mg | Sarilumab 200 mg/Sarilumab 200 mg
Number analyzed (Participants) | 184 | 184
Participants
  Glucose <=3.9 mmol/L and <LLN: number analyzed (Participants) | 181 | 184
  Glucose <=3.9 mmol/L and <LLN | 10 | 8
  Glucose >=11.1 mmol/L (unfas) or >=7 mmol/L (fas): number analyzed (Participants) | 181 | 184
  Glucose >=11.1 mmol/L (unfas) or >=7 mmol/L (fas) | 17 | 12
  HbA1c >8%: number analyzed (Participants) | 178 | 179
  HbA1c >8% | 3 | 3
  Total Cholesterol >=6.2 mmol/L: number analyzed (Participants) | 181 | 184
  Total Cholesterol >=6.2 mmol/L | 52 | 88
  Total Cholesterol >=7.74 mmol/L: number analyzed (Participants) | 181 | 184
  Total Cholesterol >=7.74 mmol/L | 15 | 14
  LDL Cholesterol >=4.1 mmol/L: number analyzed (Participants) | 180 | 184
  LDL Cholesterol >=4.1 mmol/L | 35 | 59
  LDL Cholesterol >=4.9 mmol/L: number analyzed (Participants) | 180 | 184
  LDL Cholesterol >=4.9 mmol/L | 18 | 20
  Triglycerides >=4.6 mmol/L: number analyzed (Participants) | 181 | 184
  Triglycerides >=4.6 mmol/L | 4 | 8
  Triglycerides >=5.6 mmol/L: number analyzed (Participants) | 181 | 184
  Triglycerides >=5.6 mmol/L | 3 | 6

37. Secondary Outcome: OLE Period: Number of Participants With Potentially Clinically Significant Abnormalities - Metabolic Parameters
Description: Criteria for potentially clinically significant abnormalities:
  * Glucose: <=3.9 mmol/L and <LLN; >=11.1 mmol/L (unfas) or >=7 mmol/L (fas).
  * HbA1c: >8%.
  * Total cholesterol: >=6.2 mmol/L; >=7.74 mmol/L.
  * LDL cholesterol: >=4.1 mmol/L; >=4.9 mmol/L.
  * Triglycerides: >=4.6 mmol/L; >=5.6 mmol/L.
Time Frame: From end of Week 24 (Baseline of OLE Period) up to Week 300
Population: Analysis was performed on safety population (OLE Period). Here, 'number analyzed' = participants with available data for each specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | Adalimumab 40 mg/Sarilumab 200 mg | Sarilumab 200 mg/Sarilumab 200 mg
Number analyzed (Participants) | 155 | 165
Participants
  Glucose <=3.9 mmol/L and <LLN: number analyzed (Participants) | 153 | 165
  Glucose <=3.9 mmol/L and <LLN | 5 | 6
  Glucose >=11.1 mmol/L (unfas) or >=7 mmol/L (fas): number analyzed (Participants) | 153 | 165
  Glucose >=11.1 mmol/L (unfas) or >=7 mmol/L (fas) | 20 | 14
  HbA1c >8%: number analyzed (Participants) | 147 | 161
  HbA1c >8% | 2 | 2
  Total Cholesterol >=6.2 mmol/L: number analyzed (Participants) | 153 | 165
  Total Cholesterol >=6.2 mmol/L | 77 | 69
  Total Cholesterol >=7.74 mmol/L: number analyzed (Participants) | 153 | 165
  Total Cholesterol >=7.74 mmol/L | 22 | 19
  LDL Cholesterol >=4.1 mmol/L: number analyzed (Participants) | 151 | 164
  LDL Cholesterol >=4.1 mmol/L | 57 | 48
  LDL Cholesterol >=4.9 mmol/L: number analyzed (Participants) | 151 | 164
  LDL Cholesterol >=4.9 mmol/L | 25 | 16
  Triglycerides >=4.6 mmol/L: number analyzed (Participants) | 153 | 165
  Triglycerides >=4.6 mmol/L | 13 | 6
  Triglycerides >=5.6 mmol/L: number analyzed (Participants) | 153 | 165
  Triglycerides >=5.6 mmol/L | 4 | 6

38. Secondary Outcome: DB Period: Number of Participants With Different Post-baseline Categories of High-density Lipoprotein (HDL)
Description: Number of participants with different post-baseline status of HDL: < 40 mg/dL, 40 - < 60 mg/dL, >= 60 mg/dL, is reported here.
Time Frame: From Week 0 to Week 24
Population: as for outcome 34
Measure: Count of Participants; unit: Participants
Arm/Group | Adalimumab 40 mg/Sarilumab 200 mg | Sarilumab 200 mg/Sarilumab 200 mg
Number analyzed (Participants) | 181 | 184
Participants
  HDL: < 40 mg/dL | 5 | 7
  HDL: 40 - < 60 mg/dL | 57 | 45
  HDL: >=60 mg/dL | 119 | 132

39. Secondary Outcome: OLE Period: Number of Participants With Different Post-baseline Categories of High-density Lipoprotein
Description: Number of participants with different post-baseline status of HDL: < 40 mg/dL, 40 - < 60 mg/dL, >=60 mg/dL, is reported here.
Time Frame: From end of Week 24 (Baseline of OLE Period) up to Week 300
Population: as for outcome 33
Measure: Count of Participants; unit: Participants
Arm/Group | Adalimumab 40 mg/Sarilumab 200 mg | Sarilumab 200 mg/Sarilumab 200 mg
Number analyzed (Participants) | 153 | 165
Participants
  HDL: < 40 mg/dL | 7 | 5
  HDL: 40 - < 60 mg/dL | 52 | 49
  HDL: >=60 mg/dL | 94 | 111

40. Secondary Outcome: DB Period: Number of Participants With Potentially Clinically Significant Abnormalities - Renal Function
Description: Criteria for potentially clinically significant abnormalities:
  * Creatinine: >=150 micromol/L (adults); >=30% change from baseline, >=100% change from baseline.
  * Creatinine clearance: <15 mL/min; >=15 to <30 mL/min; >=30 to <60 mL/min; >=60 to <90 mL/min.
  * Blood urea nitrogen: >=17 mmol/L.
  * Uric acid: <120 micromol/L; >408 micromol/L.
Time Frame: From Week 0 to Week 24
Population: as for outcome 34
Measure: Count of Participants; unit: Participants
Arm/Group | Adalimumab 40 mg/Sarilumab 200 mg | Sarilumab 200 mg/Sarilumab 200 mg
Number analyzed (Participants) | 183 | 184
Participants
  Creatinine >=150 micromol/L (Adults) | 0 | 3
  Creatinine >=30% change from baseline | 19 | 23
  Creatinine >=100% change from baseline | 0 | 1
  Creatinine Clearance <15 mL/min | 0 | 0
  Creatinine clearance >=15 to <30 mL/min | 0 | 1
  Creatinine clearance >=30 to <60 mL/min | 21 | 22
  Creatinine clearance >=60 to <90 mL/min | 74 | 65
  Blood Urea Nitrogen >=17 mmol/L | 0 | 2
  Uric acid <120 micromol/L | 4 | 3
  Uric acid >408 micromol/L | 25 | 35

41. Secondary Outcome: OLE Period: Number of Participants With Potentially Clinically Significant Abnormalities - Renal Function
Description: as for outcome 40
Time Frame: From end of Week 24 (Baseline of OLE Period) up to Week 300
Population: as for outcome 33
Measure: Count of Participants; unit: Participants
Arm/Group | Adalimumab 40 mg/Sarilumab 200 mg | Sarilumab 200 mg/Sarilumab 200 mg
Number analyzed (Participants) | 154 | 165
Participants
  Creatinine >=150 micromol/L (Adults) | 2 | 2
  Creatinine >=30% change from baseline | 63 | 62
  Creatinine >=100% change from baseline | 5 | 1
  Creatinine Clearance <15 mL/min | 0 | 0
  Creatinine clearance >=15 to <30 mL/min | 1 | 0
  Creatinine clearance >=30 to <60 mL/min | 34 | 24
  Creatinine clearance >=60 to <90 mL/min | 66 | 81
  Blood Urea Nitrogen >=17 mmol/L | 1 | 3
  Uric acid <120 micromol/L | 2 | 3
  Uric acid >408 micromol/L | 44 | 43

42. Secondary Outcome: DB Period: Number of Participants With Potentially Clinically Significant Abnormalities - Urinalysis
Description: Criteria with potentially clinically significant urine abnormalities:
  pH: <= 4.6; pH: >= 8.0.
Time Frame: From Week 0 to Week 24
Population: as for outcome 34
Measure: Count of Participants; unit: Participants
Arm/Group | Adalimumab 40 mg/Sarilumab 200 mg | Sarilumab 200 mg/Sarilumab 200 mg
Number analyzed (Participants) | 87 | 85
Participants
  pH <= 4.6 | 0 | 0
  pH >= 8.0 | 0 | 0

43. Secondary Outcome: OLE Period: Number of Participants With Potentially Clinically Significant Abnormalities - Urinalysis
Description: Criteria with potentially clinically significant urine abnormalities:
  pH: <= 4.6; pH: >= 8.0.
Time Frame: From end of Week 24 (Baseline of OLE Period) up to Week 300
Population: as for outcome 33
Measure: Count of Participants; unit: Participants
Arm/Group | Adalimumab 40 mg/Sarilumab 200 mg | Sarilumab 200 mg/Sarilumab 200 mg
Number analyzed (Participants) | 105 | 109
Participants
  pH <= 4.6 | 0 | 0
  pH >= 8.0 | 0 | 1

44. Secondary Outcome: DB Period: Number of Participants With Potentially Clinically Significant Abnormalities - Electrolytes
Description: Criteria for potentially clinically significant abnormalities:
  * Sodium: <=129 mmol/L; >=160 mmol/L.
  * Potassium: <3 mmol/L; >=5.5 mmol/L.
  * Chloride: <80 mmol/L; >115 mmol/L.
Time Frame: From Week 0 to Week 24
Population: as for outcome 34
Measure: Count of Participants; unit: Participants
Arm/Group | Adalimumab 40 mg/Sarilumab 200 mg | Sarilumab 200 mg/Sarilumab 200 mg
Number analyzed (Participants) | 183 | 184
Participants
  Sodium <=129 mmol/L | 1 | 1
  Sodium >=160 mmol/L | 0 | 0
  Potassium <3 mmol/L | 3 | 0
  Potassium >=5.5 mmol/L | 0 | 0
  Chloride <80 mmol/L | 0 | 0
  Chloride >115 mmol/L | 0 | 1

45. Secondary Outcome: OLE Period: Number of Participants With Potentially Clinically Significant Abnormalities - Electrolytes
Description: as for outcome 44
Time Frame: From end of Week 24 (Baseline of OLE Period) up to Week 300
Population: as for outcome 33
Measure: Count of Participants; unit: Participants
Arm/Group | Adalimumab 40 mg/Sarilumab 200 mg | Sarilumab 200 mg/Sarilumab 200 mg
Number analyzed (Participants) | 154 | 165
Participants
  Sodium <=129 mmol/L | 3 | 0
  Sodium >=160 mmol/L | 0 | 0
  Potassium <3 mmol/L | 2 | 2
  Potassium >=5.5 mmol/L | 6 | 7
  Chloride <80 mmol/L | 1 | 0
  Chloride >115 mmol/L | 0 | 0

46. Secondary Outcome: DB Period: Number of Participants With Potentially Clinically Significant Electrocardiogram (ECG) Abnormalities
Description: Criteria for potentially clinically significant ECG abnormalities:
  * Heart rate (HR): <50 beats per minute (bpm); <50 bpm and DFB >=20 bpm; <40 bpm; <40 bpm and DFB >=20 bpm; <30 bpm; <30 bpm and DFB >=20 bpm; >90 bpm; >=90 bpm and increase from baseline (IFB) >=20 bpm; >100 bpm; >=100 bpm and IFB >=20 bpm; >120 bpm; >=120 bpm and IFB >=20 bpm.
  * PR Interval: >200 millisecond (ms); >200 ms and IFB >=25%; >220 ms; >220 ms and IFB >=25%; >240 ms; >240 ms and IFB >=25%.
  * QRS Interval: >110 ms; >110 ms and IFB >=25%; >120 ms; >120 ms and IFB >=25%.
  * QT Interval: >500 ms.
  * QTc Bazett (QTc B): >450 ms; >480 ms; >500 ms; IFB >30 and <=60 ms; IFB >60 ms.
  * QTc Fridericia (QTc F): >450 ms; >480 ms; >500 ms; IFB >30 and <=60 ms; IFB >60 ms.
Time Frame: From Week 0 to Week 24
Population: Analysis was performed on safety population (DB Period). Here, 'overall number of participants analyzed' = participants evaluable for this outcome measure and 'number analyzed' = participants with available data for each specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | Adalimumab 40 mg/Sarilumab 200 mg | Sarilumab 200 mg/Sarilumab 200 mg
Number analyzed (Participants) | 163 | 162
Participants
  HR <50 bpm: number analyzed (Participants) | 162 | 161
  HR <50 bpm | 4 | 5
  HR <50 bpm and DFB >=20 bpm: number analyzed (Participants) | 158 | 158
  HR <50 bpm and DFB >=20 bpm | 0 | 0
  HR <40 bpm: number analyzed (Participants) | 162 | 161
  HR <40 bpm | 0 | 0
  HR <40 bpm and DFB >=20 bpm: number analyzed (Participants) | 158 | 158
  HR <40 bpm and DFB >=20 bpm | 0 | 0
  HR <30 bpm: number analyzed (Participants) | 162 | 161
  HR <30 bpm | 0 | 0
  HR <30 bpm and DFB >=20 bpm: number analyzed (Participants) | 158 | 158
  HR <30 bpm and DFB >=20 bpm | 0 | 0
  HR >90 bpm: number analyzed (Participants) | 162 | 161
  HR >90 bpm | 11 | 2
  HR >=90 bpm and IFB >=20 bpm: number analyzed (Participants) | 158 | 158
  HR >=90 bpm and IFB >=20 bpm | 5 | 1
  HR >100 bpm: number analyzed (Participants) | 162 | 161
  HR >100 bpm | 2 | 1
  HR >=100 bpm and IFB >=20 bpm: number analyzed (Participants) | 158 | 158
  HR >=100 bpm and IFB >=20 bpm | 2 | 0
  HR >120 bpm: number analyzed (Participants) | 162 | 161
  HR >120 bpm | 0 | 0
  HR >=120 bpm and IFB >=20 bpm: number analyzed (Participants) | 158 | 158
  HR >=120 bpm and IFB >=20 bpm | 0 | 0
  PR Interval >200 ms: number analyzed (Participants) | 163 | 161
  PR Interval >200 ms | 11 | 5
  PR Interval >200 ms and IFB >=25%: number analyzed (Participants) | 159 | 158
  PR Interval >200 ms and IFB >=25% | 1 | 0
  PR Interval >220 ms: number analyzed (Participants) | 163 | 161
  PR Interval >220 ms | 4 | 1
  PR Interval >220 ms and IFB >=25%: number analyzed (Participants) | 159 | 158
  PR Interval >220 ms and IFB >=25% | 0 | 0
  PR Interval >240 ms: number analyzed (Participants) | 163 | 161
  PR Interval >240 ms | 1 | 1
  PR Interval >240 ms and IFB >=25%: number analyzed (Participants) | 159 | 158
  PR Interval >240 ms and IFB >=25% | 0 | 0
  QRS Interval >110 ms | 3 | 9
  QRS Interval >110 ms and IFB >=25%: number analyzed (Participants) | 159 | 159
  QRS Interval >110 ms and IFB >=25% | 0 | 0
  QRS Interval >120 ms | 1 | 2
  QRS Interval >120 ms and IFB >=25%: number analyzed (Participants) | 159 | 159
  QRS Interval >120 ms and IFB >=25% | 0 | 0
  QT Interval >500 ms | 0 | 1
  QTc B >450 ms | 16 | 7
  QTc B >480 ms | 2 | 0
  QTc B >500 ms | 0 | 0
  QTc B IFB >30 and <=60 ms: number analyzed (Participants) | 159 | 159
  QTc B IFB >30 and <=60 ms | 11 | 5
  QTc B IFB >60 ms: number analyzed (Participants) | 159 | 159
  QTc B IFB >60 ms | 0 | 0
  QTc F>450 ms | 7 | 5
  QTc F>480 ms | 0 | 0
  QTc F>500 ms | 0 | 0
  QTc F IFB >30 and <=60 ms: number analyzed (Participants) | 159 | 159
  QTc F IFB >30 and <=60 ms | 9 | 3
  QTc F IFB >60 ms: number analyzed (Participants) | 159 | 159
  QTc F IFB >60 ms | 0 | 0

47. Secondary Outcome: OLE Period: Number of Participants With Potentially Clinically Significant Electrocardiogram Abnormalities
Description: Criteria for potentially clinically significant ECG abnormalities:
  * HR: <50 bpm; <50 bpm and DFB >=20 bpm; <40 bpm; <40 bpm and DFB >=20 bpm; <30 bpm; <30 bpm and DFB >=20 bpm; >90 bpm; >=90 bpm and IFB >=20 bpm; >100 bpm; >=100 bpm and IFB >=20 bpm; >120 bpm; >=120 bpm and IFB >=20 bpm.
  * PR Interval: >200 ms; >200 ms and IFB >=25%; >220 ms; >220 ms and IFB >=25%; >240 ms; >240 ms and IFB >=25%.
  * QRS Interval: >110 ms; >110 ms and IFB >=25%; >120 ms; >120 ms and IFB >=25%.
  * QT Interval: >500 ms.
  * QTc B: >450 ms; >480 ms; >500 ms; IFB >30 and <=60 ms; IFB >60 ms.
  * QTc F: >450 ms; >480 ms; >500 ms; IFB >30 and <=60 ms; IFB >60 ms.
Time Frame: From end of Week 24 (Baseline of OLE Period) up to Week 300
Population: Analysis was performed on safety population (OLE Period). Here, 'overall number analyzed' = participants evaluable for this outcome measure and 'number analyzed' = participants with available data for each specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | Adalimumab 40 mg/Sarilumab 200 mg | Sarilumab 200 mg/Sarilumab 200 mg
Number analyzed (Participants) | 154 | 163
Participants
  HR <50 bpm | 10 | 19
  HR <50 bpm and DFB >=20 bpm: number analyzed (Participants) | 152 | 159
  HR <50 bpm and DFB >=20 bpm | 0 | 3
  HR <40 bpm | 1 | 1
  HR <40 bpm and DFB >=20 bpm: number analyzed (Participants) | 152 | 159
  HR <40 bpm and DFB >=20 bpm | 0 | 1
  HR <30 bpm | 0 | 0
  HR <30 bpm and DFB >=20 bpm: number analyzed (Participants) | 152 | 159
  HR <30 bpm and DFB >=20 bpm | 0 | 0
  HR >90 bpm | 16 | 11
  HR >=90 bpm and IFB >=20 bpm: number analyzed (Participants) | 152 | 159
  HR >=90 bpm and IFB >=20 bpm | 7 | 6
  HR >100 bpm | 3 | 3
  HR >=100 bpm and IFB >=20 bpm: number analyzed (Participants) | 152 | 159
  HR >=100 bpm and IFB >=20 bpm | 2 | 1
  HR >120 bpm | 0 | 0
  HR >=120 bpm and IFB >=20 bpm: number analyzed (Participants) | 152 | 159
  HR >=120 bpm and IFB >=20 bpm | 0 | 0
  PR Interval >200 ms | 17 | 14
  PR Interval >200 ms and IFB >=25%: number analyzed (Participants) | 152 | 158
  PR Interval >200 ms and IFB >=25% | 6 | 3
  PR Interval >220 ms | 8 | 6
  PR Interval >220 ms and IFB >=25%: number analyzed (Participants) | 152 | 158
  PR Interval >220 ms and IFB >=25% | 4 | 3
  PR Interval >240 ms | 2 | 2
  PR Interval >240 ms and IFB >=25%: number analyzed (Participants) | 152 | 158
  PR Interval >240 ms and IFB >=25% | 2 | 1
  QRS Interval >110 ms | 8 | 18
  QRS Interval >110 ms and IFB >=25%: number analyzed (Participants) | 152 | 159
  QRS Interval >110 ms and IFB >=25% | 2 | 1
  QRS Interval >120 ms | 3 | 7
  QRS Interval >120 ms and IFB >=25%: number analyzed (Participants) | 152 | 159
  QRS Interval >120 ms and IFB >=25% | 1 | 0
  QT Interval >500 ms | 2 | 2
  QTc B >450 ms | 35 | 33
  QTc B >480 ms | 3 | 30
  QTc B >500 ms | 1 | 1
  QTc B IFB >30 and <=60 ms: number analyzed (Participants) | 152 | 159
  QTc B IFB >30 and <=60 ms | 18 | 23
  QTc B IFB >60 ms: number analyzed (Participants) | 152 | 159
  QTc B IFB >60 ms | 3 | 2
  QTc F>450 ms | 16 | 16
  QTc F>480 ms | 3 | 2
  QTc F>500 ms | 0 | 1
  QTc F IFB >30 and <=60 ms: number analyzed (Participants) | 152 | 159
  QTc F IFB >30 and <=60 ms | 19 | 19
  QTc F IFB >60 ms: number analyzed (Participants) | 152 | 159
  QTc F IFB >60 ms | 4 | 3

48. Secondary Outcome: DB Period: Number of Participants With Potentially Clinically Significant Vital Signs Abnormalities
Description: Criteria for potentially clinically significant vital sign abnormalities:
  Systolic blood pressure (SBP) supine: <=95 mmHg and DFB>=20 mmHg; >=160 mmHg and IFB >=20 mmHg.
  Diastolic blood pressure (DBP) supine: <=45 mmHg and DFB >=10 mmHg; >=110 mmHg and IFB >=10 mmHg.
  SBP (Orthostatic): <=-20 mmHg. DBP (Orthostatic): <=-10 mmHg. HR supine: <=50 bpm and DFB >=20 bpm; >=120 bpm and IFB >=20 bpm. Weight: >=5% DFB; >=5% IFB.
Time Frame: From Week 0 to Week 24
Population: as for outcome 32
Measure: Count of Participants; unit: Participants
Arm/Group | Adalimumab 40 mg/Sarilumab 200 mg | Sarilumab 200 mg/Sarilumab 200 mg
Number analyzed (Participants) | 184 | 184
Participants
  SBP (supine) <=95 mmHg and DFB >=20 mmHg: number analyzed (Participants) | 182 | 182
  SBP (supine) <=95 mmHg and DFB >=20 mmHg | 4 | 3
  SBP (supine) >=160 mmHg and IFB >=20 mmHg: number analyzed (Participants) | 182 | 182
  SBP (supine) >=160 mmHg and IFB >=20 mmHg | 4 | 5
  DBP (supine) <=45 mmHg and DFB >=10 mmHg: number analyzed (Participants) | 182 | 182
  DBP (supine) <=45 mmHg and DFB >=10 mmHg | 1 | 1
  DBP (supine) >=110 mmHg and IFB >=10 mmHg: number analyzed (Participants) | 182 | 182
  DBP (supine) >=110 mmHg and IFB >=10 mmHg | 1 | 1
  SBP (orthostatic) <=-20 mmHg: number analyzed (Participants) | 150 | 161
  SBP (orthostatic) <=-20 mmHg | 13 | 10
  DBP (orthostatic) <=-10 mmHg: number analyzed (Participants) | 150 | 161
  DBP (orthostatic) <=-10 mmHg | 20 | 27
  HR (supine) <=50 bpm and DFB >= 20 bpm: number analyzed (Participants) | 182 | 182
  HR (supine) <=50 bpm and DFB >= 20 bpm | 2 | 1
  HR (supine) >=120 bpm and IFB >=20 bpm: number analyzed (Participants) | 182 | 182
  HR (supine) >=120 bpm and IFB >=20 bpm | 1 | 0
  Weight >=5% DFB: number analyzed (Participants) | 178 | 180
  Weight >=5% DFB | 12 | 6
  Weight >=5% IFB: number analyzed (Participants) | 178 | 180
  Weight >=5% IFB | 21 | 23

49. Secondary Outcome: OLE Period: Number of Participants With Potentially Clinically Significant Vital Signs Abnormalities
Description: Criteria for potentially clinically significant vital sign abnormalities:
  SBP supine: <=95 mmHg and DFB >=20 mmHg; >=160 mmHg and IFB >=20 mmHg. DBP supine: <=45 mmHg and DFB >=10 mmHg; >=110 mmHg and IFB >=10 mmHg. SBP (Orthostatic): <=-20 mmHg. DBP (Orthostatic): <=-10 mmHg. HR supine: <=50 bpm and DFB >=20 bpm; >=120 bpm and IFB >=20 bpm. Weight: >=5% DFB; >=5% IFB.
Time Frame: From end of Week 24 (Baseline of OLE Period) up to Week 300
Population: as for outcome 37
Measure: Count of Participants; unit: Participants
Arm/Group | Adalimumab 40 mg/Sarilumab 200 mg | Sarilumab 200 mg/Sarilumab 200 mg
Number analyzed (Participants) | 155 | 165
Participants
  SBP (supine) <=95 mmHg and DFB >=20 mmHg: number analyzed (Participants) | 154 | 164
  SBP (supine) <=95 mmHg and DFB >=20 mmHg | 3 | 9
  SBP (supine) >=160 mmHg and IFB >=20 mmHg: number analyzed (Participants) | 154 | 164
  SBP (supine) >=160 mmHg and IFB >=20 mmHg | 10 | 11
  DBP (supine) <=45 mmHg and DFB >=10 mmHg: number analyzed (Participants) | 154 | 164
  DBP (supine) <=45 mmHg and DFB >=10 mmHg | 0 | 0
  DBP (supine) >=110 mmHg and IFB >=10 mmHg: number analyzed (Participants) | 154 | 164
  DBP (supine) >=110 mmHg and IFB >=10 mmHg | 1 | 2
  SBP (orthostatic) <=-20 mmHg: number analyzed (Participants) | 150 | 162
  SBP (orthostatic) <=-20 mmHg | 24 | 32
  DBP (orthostatic) <=-10 mmHg: number analyzed (Participants) | 150 | 162
  DBP (orthostatic) <=-10 mmHg | 41 | 46
  HR (supine) <=50 bpm and DFB >= 20 bpm: number analyzed (Participants) | 154 | 164
  HR (supine) <=50 bpm and DFB >= 20 bpm | 3 | 0
  HR (supine) >=120 bpm and IFB >=20 bpm: number analyzed (Participants) | 154 | 164
  HR (supine) >=120 bpm and IFB >=20 bpm | 0 | 0
  Weight >=5% DFB: number analyzed (Participants) | 151 | 164
  Weight >=5% DFB | 44 | 51
  Weight >=5% IFB: number analyzed (Participants) | 151 | 164
  Weight >=5% IFB | 82 | 87

50. Secondary Outcome: DB Period: Number of Participants With Treatment-emergent and Treatment-boosted Anti-drug Antibody (ADA) Response
Description: Anti-drug antibody response was categorized as: Treatment emergent and Treatment-boosted. Treatment emergent ADAs was defined as a participant with no positive assay response at baseline but with a positive assay response during the TEAE period. Treatment boosted ADAs: defined as participants with a positive ADA assay response at baseline and with at least a 4-fold increase in titer compared to baseline during the TEAE period. TEAE period: time from first dose of study drug up to day before first dose of open-label treatment for participants who completed 24-week randomized/DB treatment.
Time Frame: From Week 0 to Week 24
Population: Analysis was performed on ADA population which consisted of all participants who had signed informed consent and had been allocated to a randomized treatment; received at least 1 dose or part of a dose of IMP with at least 1 post-dose, evaluable ADA sample. Data for this outcome measure was not planned to be collected and analyzed for Adalimumab 40 mg/Sarilumab 200 mg arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Sarilumab 200 mg/Sarilumab 200 mg
Number analyzed (Participants) | 184
Participants
  Treatment-emergent ADA | 13
  Treatment-boosted ADA | 0

51. Secondary Outcome: Number of Participants With Treatment-emergent and Treatment-boosted Anti-drug Antibody Response During Entire Treatment-emergent Adverse Event Period
Description: Anti-drug antibody response was categorized as: Treatment emergent and Treatment-boosted. Treatment emergent ADAs was defined as a participant with no positive assay response at baseline but with a positive assay response during the entire TEAE period. Treatment boosted ADAs: defined as participants with a positive ADA assay response at baseline and with at least a 4-fold increase in titer compared to baseline during the entire TEAE period. Entire TEAE period: last OLE dose - first DB dose date + 6 weeks (follow-up), regardless of unplanned intermittent discontinuations.
Time Frame: From Week 0 up to last dose in OLE + 6 weeks of follow-up (i.e. up to Week 306)
Population: Analysis was performed on immunogenicity population which consisted of all participants who received at least 1 dose or part of a dose of IMP with at least 1 post-dose, evaluable ADA sample.
Measure: Count of Participants; unit: Participants
Arm/Group | Adalimumab 40 mg/Sarilumab 200 mg | Sarilumab 200 mg/Sarilumab 200 mg
Number analyzed (Participants) | 150 | 163
Participants
  Treatment-emergent ADAs | 11 | 11
  Treatment-boosted ADAs | 0 | 0

52. Secondary Outcome: DB Period: Pharmacokinetics: Serum Trough (Pre-dose) Concentrations of Functional Sarilumab
Description: Data for this outcome measure was not planned to be collected and analyzed for "Adalimumab 40 mg/Sarilumab 200 mg" arm.
Time Frame: Pre-dose at Week 0 (Baseline), 2, 4, 12, 16, 20, and 24
Population: Analysis was performed on Pharmacokinetics population (DB period) which consisted of all randomized Sarilumab participants who received at least 1 dose of IMP with at least one post-dose, non-missing concentration of functional Sarilumab in serum concentration value. Here, 'number analyzed' = participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Sarilumab 200 mg/Sarilumab 200 mg
Number analyzed (Participants) | 184
nanograms per milliliter (ng/mL)
  Baseline: number analyzed (Participants) | 177
  Baseline | 0.00 (0.00)
  Week 2: number analyzed (Participants) | 176
  Week 2 | 5566.03 (4843.57)
  Week 4: number analyzed (Participants) | 167
  Week 4 | 11209.64 (8202.70)
  Week 12: number analyzed (Participants) | 152
  Week 12 | 21355.19 (14805.63)
  Week 16: number analyzed (Participants) | 155
  Week 16 | 23143.39 (16508.71)
  Week 20: number analyzed (Participants) | 152
  Week 20 | 25252.43 (17319.04)
  Week 24: number analyzed (Participants) | 148
  Week 24 | 24233.10 (17581.72)

53. Secondary Outcome: OLE Period: Pharmacokinetics: Serum Trough (Pre-dose) Concentrations of Functional Sarilumab
Time Frame: Pre-dose at Week 24 (Baseline of OLE period), 36, 48, 60, 84, 108, 132, 156, 180, 204, 228, 252, 276, 300 and 306
Population: Analysis was performed on Pharmacokinetics population (OLE period) which consisted of all participants from the randomized population who received at least 1 dose of IMP with at least one post-dose, non-missing serum sarilumab concentration. Here, 'number analyzed' = participants with available data for each specified category and '0' denotes that no participant was available for the assessment at the specified timepoint.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Adalimumab 40 mg/Sarilumab 200 mg | Sarilumab 200 mg/Sarilumab 200 mg
Number analyzed (Participants) | 150 | 163
ng/mL
  Week 24 (Baseline of OLE period): number analyzed (Participants) | 128 | 146
  Week 24 (Baseline of OLE period) | 109.38 (1237.44) | 24403.72 (17588.31)
  Week 36: number analyzed (Participants) | 134 | 146
  Week 36 | 18952.69 (15125.86) | 26006.07 (19194.79)
  Week 48: number analyzed (Participants) | 125 | 133
  Week 48 | 21911.87 (17926.01) | 25571.16 (18958.00)
  Week 60: number analyzed (Participants) | 121 | 127
  Week 60 | 21583.82 (17594.87) | 24005.78 (18541.46)
  Week 84: number analyzed (Participants) | 104 | 108
  Week 84 | 23230.92 (18274.09) | 23873.23 (19794.57)
  Week 108: number analyzed (Participants) | 109 | 119
  Week 108 | 20405.02 (15553.02) | 21023.55 (17792.89)
  Week 132: number analyzed (Participants) | 104 | 110
  Week 132 | 20814.89 (17848.70) | 20021.53 (18580.91)
  Week 156: number analyzed (Participants) | 97 | 113
  Week 156 | 23604.11 (19660.31) | 22423.29 (18757.11)
  Week 180: number analyzed (Participants) | 96 | 105
  Week 180 | 18611.01 (16417.46) | 21856.85 (18612.43)
  Week 204: number analyzed (Participants) | 93 | 107
  Week 204 | 17982.66 (16640.61) | 18244.96 (16383.47)
  Week 228: number analyzed (Participants) | 84 | 85
  Week 228 | 19451.40 (17694.09) | 18315.19 (17525.62)
  Week 252: number analyzed (Participants) | 55 | 61
  Week 252 | 19663.10 (16020.11) | 19224.47 (16964.41)
  Week 276: number analyzed (Participants) | 52 | 63
  Week 276 | 19071.00 (18425.13) | 17014.75 (16207.18)
  Week 300: number analyzed (Participants) | 0 | 2
  Week 300 |  | 9260.00 (8683.27)
  Week 306 (Follow-up): number analyzed (Participants) | 72 | 86
  Week 306 (Follow-up) | 1237.01 (2856.88) | 2280.98 (7909.71)

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) were collected from up to Week 24 in DB period and from end of Week 24 (Baseline of OLE Period) up to Week 306 in OLE Period regardless of seriousness or relationship to study drug.
Description: Reported AEs are treatment-emergent AEs developed/worsened during 'on treatment period' (DB: time from first dose of study drug up to day before first dose of open-label treatment; OLE: from end of Week 24 [Baseline of OLE Period] up to last dose in OLE + 6 weeks [follow-up]). Analyzed on Safety population. For OLE, data was reported for pooled population (all participants received Sarilumab).
Groups:
- DB Period - Adalimumab 40 mg: Adalimumab 40 mg SC injection in combination with placebo for sarilumab q2w for 24 weeks during DB period. The dosing frequency of adalimumab was adjusted to 40 mg qw dosing in case of participants with inadequate response (<20% improvement from baseline in TJC and SJC for 2 consecutive visits) at or after Week 16 until Week 23.
- DB Period - Sarilumab 200 mg: Sarilumab 200 mg SC injection in combination with placebo for adalimumab q2w for 24 weeks during DB period. The dosing frequency of placebo for adalimumab was adjusted to 40 mg qw dosing in case of participants with inadequate response (<20% improvement from baseline in TJC and SJC for 2 consecutive visits) at or after Week 16 until Week 23.
- OLE Period - Sarilumab 200 mg: All participants who completed 24 weeks DB period had the option to continue in OLE period and received sarilumab 200 mg q2w until commercial availability of sarilumab in their country or up to maximum of additional 276 weeks (i.e. up to Week 300).
Arm/Group | DB Period - Adalimumab 40 mg | DB Period - Sarilumab 200 mg | OLE Period - Sarilumab 200 mg
All-Cause Mortality (participants affected / at risk) | 0/184 | 1/184 | 8/320
Serious Adverse Events (participants affected / at risk) | 13/184 | 9/184 | 56/320
Other Adverse Events (participants affected / at risk) | 62/184 | 79/184 | 220/320
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DB Period - Adalimumab 40 mg (N=184) | DB Period - Sarilumab 200 mg (N=184) | OLE Period - Sarilumab 200 mg (N=320)
Arthritis bacterial (Infections and infestations) | 1 | 0 | 0
Bone abscess (Infections and infestations) | 0 | 0 | 1
Bullous erysipelas (Infections and infestations) | 0 | 0 | 1
Bursitis infective (Infections and infestations) | 0 | 1 | 0
Epididymitis (Infections and infestations) | 0 | 0 | 1
Erysipelas (Infections and infestations) | 0 | 0 | 1
Mastitis (Infections and infestations) | 0 | 1 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 1
Peritonitis (Infections and infestations) | 0 | 0 | 1
Pharyngotonsillitis (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 5
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Vestibular neuronitis (Infections and infestations) | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lung adenocarcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lung squamous cell carcinoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Malignant mesenteric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Ureteric cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Yolk sac tumour site unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 2
Blood loss anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Serum sickness (Immune system disorders) | 1 | 0 | 0
Thyroid mass (Endocrine disorders) | 0 | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 1
Demyelinating polyneuropathy (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 1
Intracranial aneurysm (Nervous system disorders) | 0 | 0 | 1
Multiple sclerosis (Nervous system disorders) | 1 | 0 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 1 | 0 | 1
Cataract (Eye disorders) | 0 | 0 | 2
Uveitis (Eye disorders) | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Atrial flutter (Cardiac disorders) | 0 | 0 | 1
Cardiac failure acute (Cardiac disorders) | 0 | 1 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1
Papillary muscle rupture (Cardiac disorders) | 0 | 1 | 0
Sinus node dysfunction (Cardiac disorders) | 0 | 0 | 1
Aortic dissection (Vascular disorders) | 0 | 1 | 0
Haematoma (Vascular disorders) | 0 | 1 | 0
Iliac artery occlusion (Vascular disorders) | 0 | 0 | 1
Iliac artery stenosis (Vascular disorders) | 0 | 0 | 1
Peripheral ischaemia (Vascular disorders) | 0 | 0 | 1
Thrombophlebitis (Vascular disorders) | 0 | 0 | 1
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatic necrosis (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 2
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Biliary obstruction (Hepatobiliary disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 4
Cholestasis (Hepatobiliary disorders) | 0 | 0 | 1
Hepatic haematoma (Hepatobiliary disorders) | 0 | 0 | 1
Panniculitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 5
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1
Ureterolithiasis (Renal and urinary disorders) | 0 | 0 | 1
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 0 | 1
Uterovaginal prolapse (Reproductive system and breast disorders) | 0 | 0 | 1
Vaginal prolapse (Reproductive system and breast disorders) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Periorbital haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Device defective (Product Issues) | 0 | 0 | 1
Device dislocation (Product Issues) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DB Period - Adalimumab 40 mg (N=184) | DB Period - Sarilumab 200 mg (N=184) | OLE Period - Sarilumab 200 mg (N=320)
Bronchitis (Infections and infestations) | 7 | 12 | 41
Nasopharyngitis (Infections and infestations) | 14 | 11 | 60
Upper respiratory tract infection (Infections and infestations) | 7 | 3 | 36
Urinary tract infection (Infections and infestations) | 4 | 5 | 30
Neutropenia (Blood and lymphatic system disorders) | 1 | 25 | 59
Headache (Nervous system disorders) | 12 | 7 | 17
Hypertension (Vascular disorders) | 3 | 4 | 28
Diarrhoea (Gastrointestinal disorders) | 6 | 5 | 20
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 3 | 21
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 7 | 3 | 21
Injection site erythema (General disorders) | 7 | 14 | 26
Alanine aminotransferase increased (Investigations) | 6 | 7 | 23
Accidental overdose (Injury, poisoning and procedural complications) | 11 | 5 | 39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.